CLINICAL TRIAL: NCT03269136
Title: MAGNETISMM-1 A PHASE I, OPEN LABEL STUDY TO EVALUATE THE SAFETY, PHARMACOKINETIC, PHARMACODYNAMIC AND CLINICAL ACTIVITY OF ELRANATAMAB (PF-06863135), A B-CELL MATURATION ANTIGEN (BCMA) - CD3 BISPECIFIC ANTIBODY, AS A SINGLE AGENT AND IN COMBINATION WITH IMMUNOMODULATORY AGENTS IN PATIENTS WITH RELAPSED/REFRACTORY ADVANCED MULTIPLE MYELOMA (MM)
Brief Title: PF-06863135 As Single Agent And In Combination With Immunomodulatory Agents In Relapse/Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C1071001; 2019-000822-24 (EudraCT Number)
Record Dates: First submitted 2017-08-16; First posted 2017-08-31 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; relapse/ refractory multiple myeloma; bispecific antibody; bispecific; BCMA; BCMA- CD3 bispecific; Phase 1; PF-06863135; dexamethasone; lenalidomide; pomalidomide
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone; Lenalidomide; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- PF-06863135 (Experimental): BCMA-CD3 bispecific antibody
  Interventions: Drug: PF-06863135 monotherapy IV or SC
- PF-06863135 + dexamethasone (Experimental): BCMA-CD3 bispecific antibody + dexamethasone
  Interventions: Drug: PF-06863135 + dexamethasone
- PF-06863135 + lenalidomide (Experimental): BCMA-CD3 bispecific antibody + lenalidomide
  Interventions: Drug: PF-06863135 + lenalidomide
- PF-06863135 + pomalidomide (Experimental): BCMA-CD3 bispecific antibody + pomalidomide
  Interventions: Drug: PF-06863135 + pomalidomide

INTERVENTIONS:
Drug: PF-06863135 monotherapy IV or SC — PF-06863135 will be administered intravenously or subcutaneously.
  Other Names: BCMA-CD3 bispecific antibody
  Arms: PF-06863135
Drug: PF-06863135 + dexamethasone — PF-06863135 will be administered intravenously or subcutaneously and dexamethasone orally.
  Other Names: BCMA-CD3 bispecific antibody + dexamethasone
  Arms: PF-06863135 + dexamethasone
Drug: PF-06863135 + lenalidomide — PF-06863135 will be administered intravenously or subcutaneously and lenalidomide orally
  Other Names: BCMA-CD3 bispecific antibody + lenalidomide
  Arms: PF-06863135 + lenalidomide
Drug: PF-06863135 + pomalidomide — PF-06863135 will be administered intravenously or subcutaneously and pomalidomide orally
  Other Names: BCMA-CD3 bispecific antibody + pomalidomide
  Arms: PF-06863135 + pomalidomide

SUMMARY:
To assess the safety and tolerability at increasing dose levels of PF-06863135 in patients with relapse/ refractory multiple myeloma in order to determine the maximum tolerated dose and select the recommended Phase 2 dose.

DETAILED DESCRIPTION:
Study C1071001 is a Phase 1, open label, multi dose, multi center, dose escalation, safety, pharmacokinetic (PK) and pharmacodynamic study of PF-06863135 in adult patients with advanced multiple myeloma who have relapsed from or are refractory to standard therapy. This is a two part study; Part 1 will assess the safety and tolerability of increasing dose levels of PF-06863135 and Part 2 will evaluate safety and anti-myeloma activity of PF-06863135 at the RP2Ds determined in Part 1.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed/refractory multiple myeloma
* Progressed or are intolerant of established therapies including proteasome inhibitor, immunomodulatory drug, and anti-CD38 antibody
* Performance Status of 0- 1 ( Performance Score 2 is permitted only if due to underlying myeloma)
* Adequate bone marrow, hematological, kidney and liver function
* Resolved acute effects of any prior therapy to baseline severity
* Not pregnant

Exclusion Criteria:

* Recent history of other malignancies
* History of active autoimmune disorders
* Any form of primary immunodeficiency
* Active and clinically significant bacterial, fungal, or viral infection
* Evidence of active mucosal or internal bleeding
* History of severe immune-mediated adverse event with prior immunomodulatory treatment
* Major surgery within 4 weeks of study treatment start
* Radiation therapy within 2 weeks of study treatment start
* History of stem cell transplant (autologous or allogeneic) within 100 days prior to study enrollment
* Donor Lymphocyte Infusion (DLI) within 30 days prior to study entry
* Less than 30 days since last dose of antibody based therapies or less than 5 half-lives since last dose of previous therapy
* Requirement for systemic immune suppressive medication except as permitted in the protocol
* Current requirement for chronic blood product support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (37):
- United States (32):
  - UCSD Medical Center - Encinitas, Encinitas, California
  - UC San Diego Medical Center - La Jolla (Jacobs Medical Center / Thornton Hospital), La Jolla, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - UCSD Medical Center - Vista, Vista, California
  - Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - UChicago Medicine - River East, Chicago, Illinois
  - The University of Chicago Medical Center, CCD - Investigational Drug Service Pharmacy, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - UChicago Medicine at Ingalls - Flossmoor, Flossmoor, Illinois
  - UChicago Medicine Ingalls Memorial, Harvey, Illinois
  - University of Chicago Comprehensive Cancer Center at Silver Cross Hospital, New Lenox, Illinois
  - The University of Chicago Medicine Center for Advanced Care Orland Park, Orland Park, Illinois
  - UChicago Medicine at Ingalls - Tinley Park, Tinley Park, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center at Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center at Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center at Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center at Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center - David H. Koch Center for Cancer Care, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center at Nassau, Uniondale, New York
  - Duke University Health System: Adult Bone Marrow Transplant Clinic, Durham, North Carolina
  - Duke Cancer Center, Durham, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - Henry Joyce Cancer Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Investigational Drug Services, Baylor University Medical Center, Dallas, Texas
- Canada (5):
  - Unit 57, Special Services Building, Calgary, Alberta
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - University Health Network - Princess Margaret Cancer Centre, Toronto, Ontario
  - MUHC, GLEN site, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Lon HK, Hibma J, Jiang S, Sullivan S, Vandendries E, Skoura A, Wang D, Elmeliegy M. Population Exposure-Response Efficacy Analysis of Elranatamab (PF-06863135) in Patients with Multiple Myeloma. Target Oncol. 2025 Sep;20(5):803-819. doi: 10.1007/s11523-025-01168-y. Epub 2025 Aug 18. PMID 40826257
- [Derived] Elmeliegy M, Viqueira A, Vandendries E, Hickman A, Conte U, Irby D, Hibma J, Lon HK, Piscitelli J, Soltantabar P, Skoura A, Jiang S, Wang D. Dose Optimization of Elranatamab to Mitigate the Risk of Cytokine Release Syndrome in Patients with Multiple Myeloma. Target Oncol. 2025 Mar;20(2):349-359. doi: 10.1007/s11523-025-01134-8. Epub 2025 Feb 25. PMID 40000533
- [Derived] Bahlis NJ, Costello CL, Raje NS, Levy MY, Dholaria B, Solh M, Tomasson MH, Damore MA, Jiang S, Basu C, Skoura A, Chan EM, Trudel S, Jakubowiak A, Gasparetto C, Chu MP, Dalovisio A, Sebag M, Lesokhin AM. Elranatamab in relapsed or refractory multiple myeloma: the MagnetisMM-1 phase 1 trial. Nat Med. 2023 Oct;29(10):2570-2576. doi: 10.1038/s41591-023-02589-w. Epub 2023 Oct 2. PMID 37783970
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C1071001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 101 participants (Part 1: 86 participants and Part 2: 15 participants) were enrolled in the study.
Pre-assignment Details: The following parts were planned for the study: Part 1 dose escalation included Part 1 monotherapy, Part 1.1 dose priming, Part 1C lenalidomide combination, Part 1D pomalidomide combination and Part 1E dexamethasone combination. Part 2 dose expansion included Part 2A monotherapy, Part 2C lenalidomide combination, Part 2D pomalidomide combination and Part 2E dexamethasone combination. Participants were not enrolled in Parts 1E, 2C, 2D and 2E and their data is not reported in the record.
Groups:
- Part 1: PF-06863135 0.1 mcg/kg IV: Participants with relapsed/refractory advanced multiple myeloma (MM) received PF-06863135 at a dose of 0.1 microgram/kilogram (mcg/kg) as an intravenous (IV) infusion for 2 hours on Day 1, 8 and 15 of each 21-day cycle. Participants received treatment until disease progression, unacceptable toxicity, withdrawal of consent, death, or study termination, whichever occurred first.
- Part 1: PF-06863135 0.3 mcg/kg IV: Participants with relapsed/refractory advanced MM received PF-06863135 at a dose of 0.3 mcg/kg as an IV infusion for 2 hours on Day 1, 8 and 15 of each 21-day cycle. Participants received treatment until disease progression, unacceptable toxicity, withdrawal of consent, death, or study termination, whichever occurred first.
- Part 1: PF-06863135 1 mcg/kg IV: Participants with relapsed/refractory advanced MM received PF-06863135 at a dose of 1 mcg/kg as an IV infusion for 2 hours on Day 1, 8 and 15 of each 21-day cycle. Participants received treatment until disease progression, unacceptable toxicity, withdrawal of consent, death, or study termination, whichever occurred first.
- Part 1: PF-06863135 3 mcg/kg IV: Participants with relapsed/refractory advanced MM received PF-06863135 at a dose of 3 mcg/kg as an IV infusion for 2 hours on Day 1, 8 and 15 of each 21-day cycle. Participants received treatment until disease progression, unacceptable toxicity, withdrawal of consent, death, or study termination, whichever occurred first.
- Part 1: PF-06863135 10 mcg/kg IV: Participants with relapsed/refractory advanced MM received PF-06863135 at a dose of 10 mcg/kg as an IV infusion for 2 hours on Day 1, 8 and 15 of each 21-day cycle. Participants received treatment until disease progression, unacceptable toxicity, withdrawal of consent, death, or study termination, whichever occurred first.
- Part 1: PF-06863135 30 mcg/kg IV: Participants with relapsed/refractory advanced MM received PF-06863135 at a dose of 30 mcg/kg as an IV infusion for 2 hours on Day 1, 8 and 15 of each 21-day cycle. Participants received treatment until disease progression, unacceptable toxicity, withdrawal of consent, death, or study termination, whichever occurred first.
- Part 1: PF-06863135 50 mcg/kg IV: Participants with relapsed/refractory advanced MM received PF-06863135 at a dose of 50 mcg/kg as an IV infusion for 2 hours on Day 1, 8 and 15 of each 21-day cycle. Participants received treatment until disease progression, unacceptable toxicity, withdrawal of consent, death, or study termination, whichever occurred first.
- Part 1: PF-06863135 80 mcg/kg SC: Participants with relapsed/refractory advanced MM received PF-06863135 at a dose of 80 mcg/kg as a subcutaneous (SC) injection on Day 1, 8 and 15 of each 21-day cycle. Participants received treatment until disease progression, unacceptable toxicity, withdrawal of consent, death, or study termination, whichever occurred first.
- Part 1: PF-06863135 130 mcg/kg SC: Participants with relapsed/refractory advanced MM received PF-06863135 at a dose of 130 mcg/kg as a SC injection on Day 1, 8 and 15 of each 21-day cycle. Participants received treatment until disease progression, unacceptable toxicity, withdrawal of consent, death, or study termination, whichever occurred first.
- Part 1: PF-06863135 215 mcg/kg SC: Participants with relapsed/refractory advanced MM received PF-06863135 at a dose of 215 mcg/kg as a SC injection on Day 1, 8 and 15 of each 21-day cycle. Participants received treatment until disease progression, unacceptable toxicity, withdrawal of consent, death, or study termination, whichever occurred first.
- Part 1: PF-06863135 360 mcg/kg SC: Participants with relapsed/refractory advanced MM received PF-06863135 at a dose of 360 mcg/kg as a SC injection on Day 1, 8 and 15 of each 21-day cycle. Participants received treatment until disease progression, unacceptable toxicity, withdrawal of consent, death, or study termination, whichever occurred first.
- Part 1: PF-06863135 600 mcg/kg SC: Participants with relapsed/refractory advanced MM received PF-06863135 at a dose of 600 mcg/kg as a SC injection on Day 1, 8 and 15 of each 21-day cycle. Participants received treatment until disease progression, unacceptable toxicity, withdrawal of consent, death, or study termination, whichever occurred first.
- Part 1: PF-06863135 1000 mcg/kg SC: Participants with relapsed/refractory advanced MM received PF-06863135 at a dose of 1000 mcg/kg as a SC injection on Day 1, 8 and 15 of each 21-day cycle. Participants received treatment until disease progression, unacceptable toxicity, withdrawal of consent, death, or study termination, whichever occurred first.
- Part 1.1: PF-06863135 Priming Cohort Q1W SC: Participants with relapsed/refractory advanced MM received PF-06863135 at a priming dose of 600 mcg/kg as a SC injection, on Day 1 of Cycle 0. Participants received maintenance dose of 1000 mcg/kg as a SC injection every week (Q1W) on Day 1, 8, 15 and 22 of each 28-day cycle. Participants received treatment until disease progression, unacceptable toxicity, withdrawal of consent, death, or study termination, whichever occurred first.
- Part 1.1: PF-06863135 Priming Cohort Q2W SC: Participants with relapsed/refractory advanced MM received PF-06863135 at a priming dose of 600 mcg/kg as a SC injection, on Day 1 of Cycle 0. Participants received maintenance dose of 1000 mcg/kg as a SC injection every 2 weeks (Q2W) on Day 1 and 15 of each 28-day cycle. Participants received treatment until disease progression, unacceptable toxicity, withdrawal of consent, death, or study termination, whichever occurred first.
- Part 1C: PF-06863135 + Lenalidomide SC: Participants with relapsed/refractory advanced MM received PF-06863135 at a priming dose of 32 mcg as a SC injection, on Day 1 of Cycle 0. Participants received maintenance dose of 44 mcg as a SC injection Q1W on Day 1, 8, 15 and 22 along with lenalidomide at dose of 15 mg, orally, daily on Days 1-21 of each 28-day cycle. Participants received treatment until disease progression, unacceptable toxicity, withdrawal of consent, death, or study termination, whichever occurred first.
- Part 1D: PF-06863135 + Pomalidomide SC: Participants with relapsed/refractory advanced MM received PF-06863135 at a priming dose of 32 mcg as a SC injection, on Day 1 of Cycle 0. Participants received maintenance dose of 44 mcg as a SC injection Q1W on Day 1, 8, 15 and 22 along with pomalidomide at dose of 4 mg, orally, daily on Days 1-21 of each 28-day cycle. Participants received treatment until disease progression, unacceptable toxicity, withdrawal of consent, death, or study termination, whichever occurred first.
- Part 2A: PF-06863135 SC: Participants with relapsed/refractory advanced MM received PF-06863135 at a priming dose of 44 mcg as a SC injection, on Day 1 of Cycle 0. Participants received maintenance dose of 76 mcg as a SC injection Q1W on Day 1, 8, 15 and 22 of each 28-day cycle. Participants received treatment until disease progression, unacceptable toxicity, withdrawal of consent, death, or study termination, whichever occurred first.
Period: Part 1: Dose Escalation
Arm/Group | Part 1: PF-06863135 0.1 mcg/kg IV | Part 1: PF-06863135 0.3 mcg/kg IV | Part 1: PF-06863135 1 mcg/kg IV | Part 1: PF-06863135 3 mcg/kg IV | Part 1: PF-06863135 10 mcg/kg IV | Part 1: PF-06863135 30 mcg/kg IV | Part 1: PF-06863135 50 mcg/kg IV | Part 1: PF-06863135 80 mcg/kg SC | Part 1: PF-06863135 130 mcg/kg SC | Part 1: PF-06863135 215 mcg/kg SC | Part 1: PF-06863135 360 mcg/kg SC | Part 1: PF-06863135 600 mcg/kg SC | Part 1: PF-06863135 1000 mcg/kg SC | Part 1.1: PF-06863135 Priming Cohort Q1W SC | Part 1.1: PF-06863135 Priming Cohort Q2W SC | Part 1C: PF-06863135 + Lenalidomide SC | Part 1D: PF-06863135 + Pomalidomide SC | Part 2A: PF-06863135 SC
Started | 2 | 3 | 2 | 3 | 2 | 5 | 6 | 6 | 4 | 4 | 4 | 6 | 6 | 7 | 13 | 4 | 9 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 3 | 2 | 3 | 2 | 5 | 6 | 6 | 4 | 4 | 4 | 6 | 6 | 7 | 13 | 4 | 9 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 3 | 1 | 1 | 0
Not completed — Refused Further Treatment | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Global Deterioration of Health Status | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0
Not completed — Disease Relapse | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Progressive Disease | 2 | 3 | 2 | 3 | 2 | 5 | 3 | 5 | 3 | 1 | 2 | 2 | 3 | 3 | 8 | 3 | 4 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 1 | 0
Period: Part 2A: Dose Expansion
Arm/Group | Part 1: PF-06863135 0.1 mcg/kg IV | Part 1: PF-06863135 0.3 mcg/kg IV | Part 1: PF-06863135 1 mcg/kg IV | Part 1: PF-06863135 3 mcg/kg IV | Part 1: PF-06863135 10 mcg/kg IV | Part 1: PF-06863135 30 mcg/kg IV | Part 1: PF-06863135 50 mcg/kg IV | Part 1: PF-06863135 80 mcg/kg SC | Part 1: PF-06863135 130 mcg/kg SC | Part 1: PF-06863135 215 mcg/kg SC | Part 1: PF-06863135 360 mcg/kg SC | Part 1: PF-06863135 600 mcg/kg SC | Part 1: PF-06863135 1000 mcg/kg SC | Part 1.1: PF-06863135 Priming Cohort Q1W SC | Part 1.1: PF-06863135 Priming Cohort Q2W SC | Part 1C: PF-06863135 + Lenalidomide SC | Part 1D: PF-06863135 + Pomalidomide SC | Part 2A: PF-06863135 SC
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15 (Participants in this period were enrolled in Part 2A of the study.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Refused Further Treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Disease Relapse | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 full or partial dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: PF-06863135 0.1 mcg/kg IV | Part 1: PF-06863135 0.3 mcg/kg IV | Part 1: PF-06863135 1 mcg/kg IV | Part 1: PF-06863135 3 mcg/kg IV | Part 1: PF-06863135 10 mcg/kg IV | Part 1: PF-06863135 30 mcg/kg IV | Part 1: PF-06863135 50 mcg/kg IV | Part 1: PF-06863135 80 mcg/kg SC | Part 1: PF-06863135 130 mcg/kg SC | Part 1: PF-06863135 215 mcg/kg SC | Part 1: PF-06863135 360 mcg/kg SC | Part 1: PF-06863135 600 mcg/kg SC | Part 1: PF-06863135 1000 mcg/kg SC | Part 1.1: PF-06863135 Priming Cohort Q1W SC | Part 1.1: PF-06863135 Priming Cohort Q2W SC | Part 1C: PF-06863135 + Lenalidomide SC | Part 1D: PF-06863135 + Pomalidomide SC | Part 2A: PF-06863135 SC | Total
Number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 5 | 6 | 6 | 4 | 4 | 4 | 6 | 6 | 7 | 13 | 4 | 9 | 15 | 101
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.0 (4.24) | 67.3 (4.04) | 53.0 (0.00) | 63.3 (9.24) | 54.5 (4.95) | 70.8 (14.15) | 67.0 (8.92) | 67.3 (8.73) | 63.8 (11.64) | 68.5 (9.11) | 62.0 (3.92) | 59.5 (8.31) | 58.5 (11.48) | 60.0 (12.22) | 67.4 (7.26) | 60.5 (22.49) | 58.9 (8.33) | 66.7 (9.65) | 63.7 (10.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 0 | 0 | 1 | 1 | 5 | 6 | 1 | 2 | 1 | 3 | 4 | 5 | 4 | 1 | 3 | 7 | 47
  Male | 0 | 2 | 2 | 3 | 1 | 4 | 1 | 0 | 3 | 2 | 3 | 3 | 2 | 2 | 9 | 3 | 6 | 8 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 4
  Not Hispanic or Latino | 2 | 3 | 1 | 3 | 2 | 5 | 6 | 6 | 4 | 4 | 4 | 6 | 5 | 7 | 13 | 4 | 8 | 13 | 96
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 2 | 1 | 2 | 2 | 2 | 1 | 1 | 19
  White | 1 | 2 | 1 | 1 | 0 | 4 | 6 | 6 | 3 | 2 | 2 | 4 | 4 | 5 | 10 | 2 | 8 | 10 | 71
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Drug Limiting Toxicities (DLTs) Graded According to National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) Version (v)4.03
Description: Hematological: Grade 4 neutropenia lasting >5 days; Febrile neutropenia <1000/mm^3 with a single temperature of >38.3 degree Celsius (C) or a sustained temperature of >=38 degree C for more than one hour; grade >=3 neutropenia with infection; grade 4 thrombocytopenia; grade 3 thrombocytopenia with >= Grade 2 bleeding. Non-hematological: grade 4 adverse events (AEs); Grade 3 AE lasting >=5 days despite optimal supportive care, with exception of AE attributed to cytokine release syndrome (CRS) event; grade 3 CRS, except those CRS that had a) not been maximally treated or b) improved to <=grade 1 within 48 hours; grade 4 CRS; confirmed drug-induced liver injury (DILI) meeting Hy's law criteria; grade 4 laboratory abnormalities deemed clinically significant by the investigator reported Grade 4 AE; clinically important or persistent toxicities that were not included in above criteria were also be considered a DLT following review by the investigators and the sponsor.
Time Frame: Cycle 1 (21 Days)
Population: DLT evaluable set included all participants that had experienced a DLT in the DLT observation period or received all of their planned doses of PF-06863135 in the initial DLT observation period if Q2W dosing was being evaluated or at least all but one of their planned doses of PF-0686135 if Q1W dosing was being evaluated, provided a dose was not missed due to toxicity attributed to study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: PF-06863135 Total IV: Participants with relapsed/refractory advanced MM received PF-06863135 as an IV infusion (any dose) for 2 hours on Day 1, 8 and 15 of each 21-day cycle. Participants received treatment until disease progression, unacceptable toxicity, withdrawal of consent, death, or study termination, whichever occurred first.
- Part 1: PF-06863135 Total SC: Participants with relapsed/refractory advanced MM received PF-06863135 as a SC injection (any dose) on Day 1, 8 and 15 of each 21-day cycle. Participants received treatment until disease progression, unacceptable toxicity, withdrawal of consent, death, or study termination, whichever occurred first.
- Part 1.1: PF-06863135 Total SC: Participants with relapsed/refractory advanced MM received PF-06863135 at a priming dose of 600 mcg/kg as a SC injection, on Day 1 of Cycle 0. Participants received maintenance dose of 1000 mcg/kg as a SC injection Q1W on Day 1, 8 ,15 and 22 of each 28-day cycle or Q2W on Day 1 and 15 of each 28-day cycle. Participants received treatment until disease progression, unacceptable toxicity, withdrawal of consent, death, or study termination, whichever occurred first.
Arm/Group | Part 1: PF-06863135 0.1 mcg/kg IV | Part 1: PF-06863135 0.3 mcg/kg IV | Part 1: PF-06863135 1 mcg/kg IV | Part 1: PF-06863135 3 mcg/kg IV | Part 1: PF-06863135 10 mcg/kg IV | Part 1: PF-06863135 30 mcg/kg IV | Part 1: PF-06863135 50 mcg/kg IV | Part 1: PF-06863135 80 mcg/kg SC | Part 1: PF-06863135 130 mcg/kg SC | Part 1: PF-06863135 215 mcg/kg SC | Part 1: PF-06863135 360 mcg/kg SC | Part 1: PF-06863135 600 mcg/kg SC | Part 1: PF-06863135 1000 mcg/kg SC | Part 1.1: PF-06863135 Priming Cohort Q1W SC | Part 1.1: PF-06863135 Priming Cohort Q2W SC | Part 1C: PF-06863135 + Lenalidomide SC | Part 1D: PF-06863135 + Pomalidomide SC | Part 1: PF-06863135 Total IV | Part 1: PF-06863135 Total SC | Part 1.1: PF-06863135 Total SC
Number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 5 | 6 | 6 | 4 | 4 | 4 | 6 | 6 | 5 | 9 | 2 | 6 | 23 | 30 | 14
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 2 | 0 | 1

2. Primary Outcome: Part 2: Objective Response Rate (ORR) as Per International Myeloma Working Group (IMWG) Criteria
Description: ORR per IMWG criteria: percentage of participants with best overall response (BOR) of stringent complete response (sCR), complete response (CR), very good partial response (VGPR) or partial response (PR). sCR: complete response plus normal free light chain (FLC) ratio and absence of clonal cells in bone marrow biopsy by immunohistochemistry; CR: negative immunofixation on serum and urine and disappearance of any soft tissue plasmacytomas and <5% plasma cells in bone marrow aspirates. VGPR: serum and urine M-protein detectable by immunofixation but not on electrophoresis or >=90% reduction in serum M-protein plus urine M-protein level <100 mg/24 hr. PR: >=50% reduction of serum M-protein and reduction in 24 hrs urinary M-protein by >=90% or to <200 mg/24 hr. If serum and urine M-protein were unmeasurable, >=50% decrease in difference between involved and uninvolved FLC levels required in place of the M-protein criteria.
Time Frame: From the first dose of study treatment until the first documented sCR or CR or PR or VGPR or new anti-cancer therapies or death, whichever occurred first (maximum up to 34.3 months)
Population: Modified intent to treat (mITT) analysis set included all participants who have received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 2A: PF-06863135 SC
Number analyzed (Participants) | 15
Percentage of participants | 60.0 [35.7 to 80.2]

3. Primary Outcome: Part 2: Duration of Response (DOR) as Per IMWG Criteria
Description: DOR per IMWG criteria:time from first documentation of objective tumor (OT)response to first documentation of OTprogression or to death due to any cause, whichever occurred first.sCR: CR plus normal FLC ratio & absence of clonal cells in bone marrow biopsy by immunohistochemistry;CR:Negative immunofixation on serum & urine & disappearance of any soft tissue plasmacytomas&<5% plasma cells in bone marrow aspirates.VGPR: serum & urine M-protein(Mp) detectable by immunofixation but not on electrophoresis or >=90% reduction in serum Mp plus urine Mp level <100 mg/24 hr. PR: >=50% reduction of serum Mp & reduction in 24 hrs urinary Mp by >=90% or to <200 mg/24 hr.If serum & urine Mp were unmeasurable, >=50% decrease in difference between involved & uninvolved FLC levels required in place of Mp criteria. Progression: appearance of local, regional or distant disease of same type after CR or progression of pre-existing lesions. It did not include second primary malignancies of unrelated types.
Time Frame: From the first documentation of objective tumor response to first documentation of objective tumor progression or new anti-cancer therapies or death, whichever occurred first, (maximum up to 34.3 months)
Population: mITT analysis set included all participants who have received at least one dose of study treatment. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2A: PF-06863135 SC
Number analyzed (Participants) | 9
Months | 11.6 [2.5 to NA] — The upper limit of 95% confidence interval (CI) was not estimable due to insufficient number of participants with events.

4. Secondary Outcome: Part 1: Number of Participants With Treatment Emergent Adverse Events (AEs), Serious AEs, Treatment Related AEs, Grade 3 or 4 AEs and Grade 5 AEs as Graded by NCI CTCAE v4.03
Description: AE: any untoward medical occurrence in clinical study participant, temporally associated with use of study intervention, whether or not considered related to intervention. TEAE: any event increasing in severity from baseline or event started during PF-06863135 therapy or within 30 days of last dose of drug. SAE: any untoward medical occurrence at any dose that resulted in either: death; life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect; suspected transmission via Pfizer product of infectious agent, pathogenic or non-pathogenic; or considered as important event. Treatment-related AE: AEs attributed to drug in participants who received drug. Relatedness was judged by investigator. NCI CTCAE v4.03, Grade 3= severe AE, Grade 4= life-threatening, urgent intervention indicated, Grade 5= death related to AE. AEs included SAEs and all non-SAEs.
Time Frame: From first dose of the study treatment (Day 1) up to 30 days after the last dose of study treatment (maximum up to of 43.3 months)
Population: Safety analysis set included all participants who receive at least 1 full or partial dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: PF-06863135 0.1 mcg/kg IV | Part 1: PF-06863135 0.3 mcg/kg IV | Part 1: PF-06863135 1 mcg/kg IV | Part 1: PF-06863135 3 mcg/kg IV | Part 1: PF-06863135 10 mcg/kg IV | Part 1: PF-06863135 30 mcg/kg IV | Part 1: PF-06863135 50 mcg/kg IV | Part 1: PF-06863135 80 mcg/kg SC | Part 1: PF-06863135 130 mcg/kg SC | Part 1: PF-06863135 215 mcg/kg SC | Part 1: PF-06863135 360 mcg/kg SC | Part 1: PF-06863135 600 mcg/kg SC | Part 1: PF-06863135 1000 mcg/kg SC | Part 1.1: PF-06863135 Priming Cohort Q1W SC | Part 1.1: PF-06863135 Priming Cohort Q2W SC | Part 1C: PF-06863135 + Lenalidomide SC | Part 1D: PF-06863135 + Pomalidomide SC | Part 1: PF-06863135 Total IV | Part 1: PF-06863135 Total SC | Part 1.1: PF-06863135 Total SC
Number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 5 | 6 | 6 | 4 | 4 | 4 | 6 | 6 | 7 | 13 | 4 | 9 | 23 | 30 | 20
Participants
  Participants with AEs | 2 | 3 | 2 | 3 | 2 | 5 | 6 | 6 | 4 | 4 | 4 | 6 | 6 | 7 | 13 | 4 | 9 | 23 | 30 | 20
  Participants with serious TEAEs | 0 | 1 | 0 | 3 | 0 | 2 | 5 | 4 | 1 | 3 | 3 | 4 | 5 | 6 | 9 | 2 | 8 | 11 | 20 | 15
  Participants with treatment related AEs | 2 | 1 | 1 | 1 | 2 | 4 | 6 | 4 | 4 | 4 | 4 | 6 | 6 | 7 | 13 | 4 | 9 | 17 | 28 | 20
  Participants with grade 3 or 4 AEs | 1 | 2 | 1 | 2 | 2 | 3 | 6 | 3 | 4 | 3 | 4 | 4 | 6 | 3 | 12 | 4 | 7 | 17 | 24 | 15
  Participants with grade 5 AEs | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 2 | 0 | 3 | 1 | 0 | 2 | 2 | 6 | 4

5. Secondary Outcome: Part 1: Number of Participants With Shifts From Grade Less Than or Equal to (<=) 2 at Baseline to Grade 3 or 4 Post-Baseline in Hematology Parameters
Description: Hematology parameters included: activated partial thromboplastin time prolonged, anemia, hemoglobin increased, international normalized ratio (INR) increased, leukocytosis, lymphocyte count decreased, lymphocyte count increased, neutrophil count decreased, platelet count decreased and, white blood cell decreased. According to NCI CTCAE version 4.03: Grade 1= mild, Gade 2= moderate, Grade 3= severe AE, Grade 4= life-threatening, urgent intervention indicated, Grade 5= death related to AE. In this outcome measure number of participants with shifts from grade 2 at baseline to grade 3 or 4 post-baseline in any of hematology parameters are reported.
Time Frame: as for outcome 4
Population: Safety analysis set included all participants who receive at least 1 full or partial dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: PF-06863135 0.1 mcg/kg IV | Part 1: PF-06863135 0.3 mcg/kg IV | Part 1: PF-06863135 1 mcg/kg IV | Part 1: PF-06863135 3 mcg/kg IV | Part 1: PF-06863135 10 mcg/kg IV | Part 1: PF-06863135 30 mcg/kg IV | Part 1: PF-06863135 50 mcg/kg IV | Part 1: PF-06863135 80 mcg/kg SC | Part 1: PF-06863135 130 mcg/kg SC | Part 1: PF-06863135 215 mcg/kg SC | Part 1: PF-06863135 360 mcg/kg SC | Part 1: PF-06863135 600 mcg/kg SC | Part 1: PF-06863135 1000 mcg/kg SC | Part 1.1: PF-06863135 Priming Cohort Q1W SC | Part 1.1: PF-06863135 Priming Cohort Q2W SC | Part 1C: PF-06863135 + Lenalidomide SC | Part 1D: PF-06863135 + Pomalidomide SC | Part 1: PF-06863135 Total IV | Part 1: PF-06863135 Total SC | Part 1.1: PF-06863135 Total SC
Number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 5 | 6 | 6 | 4 | 4 | 4 | 6 | 6 | 7 | 13 | 4 | 9 | 23 | 30 | 20
Participants | 1 | 2 | 2 | 2 | 2 | 5 | 5 | 6 | 3 | 4 | 4 | 6 | 6 | 6 | 13 | 4 | 9 | 19 | 29 | 19

6. Secondary Outcome: Part 1: Number of Participants With Shifts From Grade <= 2 at Baseline to Grade 3 or 4 Post-Baseline in Clinical Chemistry Parameters
Description: Clinical chemistry parameters included: alanine aminotransferase increased, alkaline phosphatase increased, aspartate aminotransferase increased, blood bilirubin increased, creatinine increased, hypercalcemia, hyperglycemia, hyperkalemia, hypermagnesemia, hypernatremia, hypoalbuminemia, hypocalcemia, hypoglycemia, hypokalemia, hypomagnesemia, hyponatremia and hypophosphatemia. According to NCI CTCAE version 4.03: Grade 1= mild, Gade 2= moderate, Grade 3= severe AE, Grade 4= life-threatening, urgent intervention indicated, Grade 5= death related to AE. In this outcome measure number of participants with shifts from grade 2 at baseline to grade 3 or 4 post-baseline in any of clinical chemistry parameters are reported.
Time Frame: as for outcome 4
Population: Safety analysis set included all participants who receive at least 1 full or partial dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: PF-06863135 0.1 mcg/kg IV | Part 1: PF-06863135 0.3 mcg/kg IV | Part 1: PF-06863135 1 mcg/kg IV | Part 1: PF-06863135 3 mcg/kg IV | Part 1: PF-06863135 10 mcg/kg IV | Part 1: PF-06863135 30 mcg/kg IV | Part 1: PF-06863135 50 mcg/kg IV | Part 1: PF-06863135 80 mcg/kg SC | Part 1: PF-06863135 130 mcg/kg SC | Part 1: PF-06863135 215 mcg/kg SC | Part 1: PF-06863135 360 mcg/kg SC | Part 1: PF-06863135 600 mcg/kg SC | Part 1: PF-06863135 1000 mcg/kg SC | Part 1.1: PF-06863135 Priming Cohort Q1W SC | Part 1.1: PF-06863135 Priming Cohort Q2W SC | Part 1C: PF-06863135 + Lenalidomide SC | Part 1D: PF-06863135 + Pomalidomide SC | Part 1: PF-06863135 Total IV | Part 1: PF-06863135 Total SC | Part 1.1: PF-06863135 Total SC
Number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 5 | 6 | 6 | 4 | 4 | 4 | 6 | 6 | 7 | 13 | 4 | 9 | 23 | 30 | 20
Participants | 0 | 2 | 0 | 1 | 0 | 2 | 1 | 2 | 0 | 2 | 2 | 3 | 2 | 3 | 8 | 4 | 3 | 6 | 11 | 11

7. Secondary Outcome: Part 1: Number of Participants With Shifts From Grade <=2 at Baseline to Grade 3 or 4 Post-Baseline in Urinalysis
Description: Proteinuria was estimated in urinalysis. According to NCI CTCAE version 4.03: Grade 1= mild, Gade 2= moderate, Grade 3= severe AE, Grade 4= life-threatening, urgent intervention indicated, Grade 5= death related to AE. In this outcome measure number of participants with shifts from grade 2 at baseline to grade 3 or 4 post-baseline in any of urinalysis parameters are reported.
Time Frame: as for outcome 4
Population: Safety analysis set included all participants who receive at least 1 full or partial dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: PF-06863135 0.1 mcg/kg IV | Part 1: PF-06863135 0.3 mcg/kg IV | Part 1: PF-06863135 1 mcg/kg IV | Part 1: PF-06863135 3 mcg/kg IV | Part 1: PF-06863135 10 mcg/kg IV | Part 1: PF-06863135 30 mcg/kg IV | Part 1: PF-06863135 50 mcg/kg IV | Part 1: PF-06863135 80 mcg/kg SC | Part 1: PF-06863135 130 mcg/kg SC | Part 1: PF-06863135 215 mcg/kg SC | Part 1: PF-06863135 360 mcg/kg SC | Part 1: PF-06863135 600 mcg/kg SC | Part 1: PF-06863135 1000 mcg/kg SC | Part 1.1: PF-06863135 Priming Cohort Q1W SC | Part 1.1: PF-06863135 Priming Cohort Q2W SC | Part 1C: PF-06863135 + Lenalidomide SC | Part 1D: PF-06863135 + Pomalidomide SC | Part 1: PF-06863135 Total IV | Part 1: PF-06863135 Total SC | Part 1.1: PF-06863135 Total SC
Number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 5 | 6 | 6 | 4 | 4 | 4 | 6 | 6 | 7 | 13 | 4 | 9 | 23 | 30 | 20
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Part 1: ORR as Per IMWG Criteria
Description: as for outcome 2
Time Frame: From the first dose of study treatment until the first documented sCR or CR or PR or VGPR or new anti-cancer therapies or death, whichever occurred first (maximum up to 63.31 months)
Population: mITT analysis set included all participants who have received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 1: PF-06863135 0.1 mcg/kg IV | Part 1: PF-06863135 0.3 mcg/kg IV | Part 1: PF-06863135 1 mcg/kg IV | Part 1: PF-06863135 3 mcg/kg IV | Part 1: PF-06863135 10 mcg/kg IV | Part 1: PF-06863135 30 mcg/kg IV | Part 1: PF-06863135 50 mcg/kg IV | Part 1: PF-06863135 80 mcg/kg SC | Part 1: PF-06863135 130 mcg/kg SC | Part 1: PF-06863135 215 mcg/kg SC | Part 1: PF-06863135 360 mcg/kg SC | Part 1: PF-06863135 600 mcg/kg SC | Part 1: PF-06863135 1000 mcg/kg SC | Part 1.1: PF-06863135 Priming Cohort Q1W SC | Part 1.1: PF-06863135 Priming Cohort Q2W SC | Part 1C: PF-06863135 + Lenalidomide SC | Part 1D: PF-06863135 + Pomalidomide SC | Part 1: PF-06863135 Total IV | Part 1: PF-06863135 Total SC | Part 1.1: PF-06863135 Total SC
Number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 5 | 6 | 6 | 4 | 4 | 4 | 6 | 6 | 7 | 13 | 4 | 9 | 23 | 30 | 20
Percentage of participants | 0 [0.0 to 65.8] | 0 [0.0 to 56.1] | 0 [0.0 to 65.8] | 0 [0.0 to 56.1] | 0 [0.0 to 65.8] | 0 [0.0 to 43.4] | 0 [0.0 to 39.0] | 0 [0.0 to 39.0] | 0 [0.0 to 49.0] | 50.0 [15.0 to 85.0] | 75.0 [30.1 to 95.4] | 66.7 [30.0 to 90.3] | 83.3 [43.6 to 97.0] | 57.1 [25.0 to 84.2] | 61.5 [25.5 to 82.3] | 75.0 [30.1 to 95.4] | 77.8 [45.3 to 93.7] | 0 [0.0 to 14.3] | 46.7 [30.2 to 63.9] | 60.0 [38.7 to 78.1]

9. Secondary Outcome: Part 1: Time to Response (TTR) as Per IMWG Criteria
Description: TTR: Defined for participants with confirmed objective response as time from first dose to first documentation of objective tumor response. sCR: complete response + normal FLC ratio & absence of clonal cells in bone marrow biopsy by immunohistochemistry; CR: Negative immunofixation on serum& urine & disappearance of soft tissue plasmacytomas & <5% plasma cells in bone marrow aspirates. VGPR: serum& urine M-protein detectable by immunofixation but not on electrophoresis or >=90% reduction in serum M-protein plus urine M-protein level <100 mg/24 hr. PR: >=50% reduction of serum M-protein& reduction in 24hrs urinary M-protein by >=90% or <200 mg/24hr. If serum & urine M-protein unmeasurable, >=50% decrease in difference between involved & uninvolved FLC levels required in place of M-protein criteria. Progression: Appearance of local, regional, distant disease of same type after CR or progression of pre-existing lesions. It didn't include second primary malignancies of unrelated types.
Time Frame: as for outcome 8
Population: mITT analysis set included all participants who have received at least one dose of study treatment. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure and for arms where it is "0" signifies there was no participant with confirmed objective response.
Measure: Median (Full Range); unit: Days
Arm/Group | Part 1: PF-06863135 0.1 mcg/kg IV | Part 1: PF-06863135 0.3 mcg/kg IV | Part 1: PF-06863135 1 mcg/kg IV | Part 1: PF-06863135 3 mcg/kg IV | Part 1: PF-06863135 10 mcg/kg IV | Part 1: PF-06863135 30 mcg/kg IV | Part 1: PF-06863135 50 mcg/kg IV | Part 1: PF-06863135 80 mcg/kg SC | Part 1: PF-06863135 130 mcg/kg SC | Part 1: PF-06863135 215 mcg/kg SC | Part 1: PF-06863135 360 mcg/kg SC | Part 1: PF-06863135 600 mcg/kg SC | Part 1: PF-06863135 1000 mcg/kg SC | Part 1.1: PF-06863135 Priming Cohort Q1W SC | Part 1.1: PF-06863135 Priming Cohort Q2W SC | Part 1C: PF-06863135 + Lenalidomide SC | Part 1D: PF-06863135 + Pomalidomide SC | Part 1: PF-06863135 Total IV | Part 1: PF-06863135 Total SC | Part 1.1: PF-06863135 Total SC
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 4 | 5 | 4 | 8 | 3 | 7 | 0 | 14 | 12
Days |  |  |  |  |  |  |  |  |  | 22.0 [22 to 22] | 22.0 [22 to 24] | 22.0 [21 to 23] | 42.0 [22 to 92] | 39.0 [8 to 65] | 36.0 [7 to 73] | 52.0 [8 to 281] | 50.0 [7 to 105] |  | 22.0 [21 to 92] | 36.0 [7 to 73]

10. Secondary Outcome: Part 1: Complete Response Rate (CRR) as Per IMWG Criteria
Description: CRR: percentage of participants with complete response (sCR or CR). sCR: complete response plus normal FLC ratio and absence of clonal cells in bone marrow biopsy by immunohistochemistry; CR: negative immunofixation on serum and urine and disappearance of any soft tissue plasmacytomas and <5% plasma cells in bone marrow aspirates.
Time Frame: From the first dose of study treatment until the first documented sCR or CR or new anti-cancer therapies or death, whichever occurred first (maximum up to 63.31 months)
Population: mITT analysis set included all participants who have received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 1: PF-06863135 0.1 mcg/kg IV | Part 1: PF-06863135 0.3 mcg/kg IV | Part 1: PF-06863135 1 mcg/kg IV | Part 1: PF-06863135 3 mcg/kg IV | Part 1: PF-06863135 10 mcg/kg IV | Part 1: PF-06863135 30 mcg/kg IV | Part 1: PF-06863135 50 mcg/kg IV | Part 1: PF-06863135 80 mcg/kg SC | Part 1: PF-06863135 130 mcg/kg SC | Part 1: PF-06863135 215 mcg/kg SC | Part 1: PF-06863135 360 mcg/kg SC | Part 1: PF-06863135 600 mcg/kg SC | Part 1: PF-06863135 1000 mcg/kg SC | Part 1.1: PF-06863135 Priming Cohort Q1W SC | Part 1.1: PF-06863135 Priming Cohort Q2W SC | Part 1C: PF-06863135 + Lenalidomide SC | Part 1D: PF-06863135 + Pomalidomide SC | Part 1: PF-06863135 Total IV | Part 1: PF-06863135 Total SC | Part 1.1: PF-06863135 Total SC
Number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 5 | 6 | 6 | 4 | 4 | 4 | 6 | 6 | 7 | 13 | 4 | 9 | 23 | 30 | 20
Percentage of participants | 0 [0.0 to 65.8] | 0 [0.0 to 56.1] | 0 [0.0 to 65.8] | 0 [0.0 to 56.1] | 0 [0.0 to 65.8] | 0 [0.0 to 43.4] | 0 [0.0 to 39.0] | 0 [0.0 to 39.0] | 0 [0.0 to 49.0] | 50.0 [15.0 to 85.0] | 25.0 [4.6 to 69.9] | 50.0 [18.8 to 81.2] | 50.0 [18.8 to 81.2] | 14.3 [2.6 to 51.3] | 46.2 [23.2 to 70.9] | 50.0 [15.0 to 85.0] | 33.3 [12.1 to 64.6] | 0 [0.0 to 14.3] | 30.0 [16.7 to 47.9] | 35.0 [18.1 to 56.7]

11. Secondary Outcome: Part 1: DOR as Per IMWG Criteria
Description: as for outcome 3
Time Frame: From the first documentation of objective tumor response to first documentation of objective tumor progression or new anti-cancer therapies or death, whichever occurred first, (maximum up to 63.31 months)
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1: PF-06863135 0.1 mcg/kg IV | Part 1: PF-06863135 0.3 mcg/kg IV | Part 1: PF-06863135 1 mcg/kg IV | Part 1: PF-06863135 3 mcg/kg IV | Part 1: PF-06863135 10 mcg/kg IV | Part 1: PF-06863135 30 mcg/kg IV | Part 1: PF-06863135 50 mcg/kg IV | Part 1: PF-06863135 80 mcg/kg SC | Part 1: PF-06863135 130 mcg/kg SC | Part 1: PF-06863135 215 mcg/kg SC | Part 1: PF-06863135 360 mcg/kg SC | Part 1: PF-06863135 600 mcg/kg SC | Part 1: PF-06863135 1000 mcg/kg SC | Part 1.1: PF-06863135 Priming Cohort Q1W SC | Part 1.1: PF-06863135 Priming Cohort Q2W SC | Part 1C: PF-06863135 + Lenalidomide SC | Part 1D: PF-06863135 + Pomalidomide SC | Part 1: PF-06863135 Total IV | Part 1: PF-06863135 Total SC | Part 1.1: PF-06863135 Total SC
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 4 | 5 | 4 | 8 | 3 | 7 | 0 | 14 | 12
Months |  |  |  |  |  |  |  |  |  | 25.3 [18.4 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 13.6 [5.4 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | NA [32.2 to NA] — The median and upper limit of 95% CI was not estimable due to insufficient number of participants with events. | NA [6.3 to NA] — The median and upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 6.7 [3.7 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 17.1 [10.6 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 14.9 [11.8 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 8.3 [2.9 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. |  | 32.2 [7.0 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 13.3 [6.3 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events.

12. Secondary Outcome: Part 1: Duration of Complete Response (DoCR) as Per IMWG Criteria
Description: DoCR was defined for participants with confirmed complete response (sCR or CR) as the time from the first documentation of complete response to the first documentation of objective tumor progression or to death due to any cause, whichever occurred first. sCR: complete response plus normal FLC ratio and absence of clonal cells in bone marrow biopsy by immunohistochemistry; CR: Negative immunofixation on serum and urine and disappearance of any soft tissue plasmacytomas and <5% plasma cells in bone marrow aspirates. Progression was defined as appearance of local, regional or distant disease of same type after CR or progression of pre-existing lesions. It didn't include second primary malignancies of unrelated types.
Time Frame: From the first documentation of complete response to the first documentation of tumor progression or death, whichever occurred first (maximum up to 63.31 months)
Population: mITT analysis set included all participants who have received at least one dose of study treatment. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure and for arms where it is "0" signifies there was no participant with complete response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1: PF-06863135 0.1 mcg/kg IV | Part 1: PF-06863135 0.3 mcg/kg IV | Part 1: PF-06863135 1 mcg/kg IV | Part 1: PF-06863135 3 mcg/kg IV | Part 1: PF-06863135 10 mcg/kg IV | Part 1: PF-06863135 30 mcg/kg IV | Part 1: PF-06863135 50 mcg/kg IV | Part 1: PF-06863135 80 mcg/kg SC | Part 1: PF-06863135 130 mcg/kg SC | Part 1: PF-06863135 215 mcg/kg SC | Part 1: PF-06863135 360 mcg/kg SC | Part 1: PF-06863135 600 mcg/kg SC | Part 1: PF-06863135 1000 mcg/kg SC | Part 1.1: PF-06863135 Priming Cohort Q1W SC | Part 1.1: PF-06863135 Priming Cohort Q2W SC | Part 1C: PF-06863135 + Lenalidomide SC | Part 1D: PF-06863135 + Pomalidomide SC | Part 1: PF-06863135 Total IV | Part 1: PF-06863135 Total SC | Part 1.1: PF-06863135 Total SC
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 3 | 1 | 6 | 2 | 3 | 0 | 9 | 9
Months |  |  |  |  |  |  |  |  |  | 25.3 [18.4 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | NA [NA to NA] — Median and CI could not be reported as participant did not have event. | NA [NA to NA] — Only one participant had event, hence median and CI not reported. Individual participant data was 31.5 months. | NA [7.0 to NA] — The median and upper limit of 95% CI was not estimable due to insufficient number of participants with events. | NA [NA to NA] — Only one participant was evaluable and had event, hence median and CI not reported. Individual participant data was 1.9 months. | NA [6.5 to NA] — The median and upper limit of 95% CI was not estimable due to insufficient number of participants with events | NA [10.3 to NA] — The median and upper limit of 95% CI was not estimable due to insufficient number of participants with events. | NA [3.7 to NA] — The median and upper limit of 95% CI was not estimable due to insufficient number of participants with events. |  | 31.5 [7.0 to NA] — The upper limit of 95% CI was not estimable due to low number of participants with events. | 11.5 [1.9 to NA] — The upper limit of 95% CI was not estimable due to low number of participants with events.

13. Secondary Outcome: Part 1: Duration of Stable Disease (DOSD) as Per IMWG Criteria
Description: DOSD per IMWG criteria: participants with confirmed stable disease (SD): time from first documentation (doc) of objective SD to first doc of objective tumor progression (P)/death by any cause, whichever occurred first. SD: not meeting criteria for CR,VGPR, PR, MR or PD. CR: Negative immunofixation on serum & urine &disappearance of any soft tissue plasmacytomas &<5% plasma cells in bone marrow aspirates. VGPR: serum & urine M-protein (Mp) detectable by immunofixation but not on electrophoresis or >=90% reduction in serum Mp plus urine Mp level <100 mg/24 hr. PR: >=50% reduction of serum Mp & reduction in 24 hours urinary Mp by >=90% or<200 mg/24 hr. If serum & urine Mp were unmeasurable, >=50% decrease in difference between involved & uninvolved FLC levels required in place of Mp criteria. Progression: appearance of local, regional, distant disease of same type after CR or progression of pre-existing lesions. It didn't include second primary malignancies of unrelated types.
Time Frame: Time from the first documentation of objective stable disease to the first documentation of objective tumor progression or to death due to any cause, whichever occurred first (maximum up to 63.31 months)
Population: mITT analysis set included all participants who have received at least one dose of study treatment. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure and for arm where it is "0" signifies there was no participant with stable disease.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1: PF-06863135 0.1 mcg/kg IV | Part 1: PF-06863135 0.3 mcg/kg IV | Part 1: PF-06863135 1 mcg/kg IV | Part 1: PF-06863135 3 mcg/kg IV | Part 1: PF-06863135 10 mcg/kg IV | Part 1: PF-06863135 30 mcg/kg IV | Part 1: PF-06863135 50 mcg/kg IV | Part 1: PF-06863135 80 mcg/kg SC | Part 1: PF-06863135 130 mcg/kg SC | Part 1: PF-06863135 215 mcg/kg SC | Part 1: PF-06863135 360 mcg/kg SC | Part 1: PF-06863135 600 mcg/kg SC | Part 1: PF-06863135 1000 mcg/kg SC | Part 1.1: PF-06863135 Priming Cohort Q1W SC | Part 1.1: PF-06863135 Priming Cohort Q2W SC | Part 1C: PF-06863135 + Lenalidomide SC | Part 1D: PF-06863135 + Pomalidomide SC | Part 1: PF-06863135 Total IV | Part 1: PF-06863135 Total SC | Part 1.1: PF-06863135 Total SC
Number analyzed (Participants) | 0 | 2 | 1 | 2 | 1 | 3 | 4 | 4 | 2 | 4 | 3 | 5 | 5 | 6 | 9 | 4 | 9 | 13 | 23 | 15
Months |  | 1.3 [0.5 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | NA [NA to NA] — Only one participant was evaluable and had event, hence median and CI not reported. Individual participant data was 0.7 months. | 0.8 [0.6 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | NA [NA to NA] — Only one participant was evaluable and had event, hence median and CI not reported. Individual participant data was 1.8 months. | 3.4 [1.0 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 3.0 [2.2 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 0.4 [0.3 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 0.6 [0.5 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 18.4 [4.2 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 13.6 [5.4 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 32.2 [2.1 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | NA [7.0 to NA] — The median and upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 7.4 [3.7 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 17.6 [11.5 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 17.9 [1.5 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 5.6 [0.7 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 1.8 [0.6 to 3.4] | 7.3 [1.4 to 32.3] | 12.0 [7.4 to 20.2]

14. Secondary Outcome: Part 1: Progression Free Survival (PFS) as Per IMWG Criteria
Description: PFS as per IMWG criteria was the time from start date of study treatment to date of first documentation of progression, or death due to any cause. Progression was defined as the appearance of local, regional or distant disease of the same type after CR or progression of pre-existing lesions. It does not include second primary malignancies of unrelated types. CR: Negative immunofixation on serum and urine and disappearance of any soft tissue plasmacytomas and <5% plasma cells in bone marrow aspirates.
Time Frame: From start date of study treatment to date of first documentation of progression or death due to any cause, whichever occurred first (maximum up to 63.31 months)
Population: mITT analysis set included all participants who have received at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1: PF-06863135 0.1 mcg/kg IV | Part 1: PF-06863135 0.3 mcg/kg IV | Part 1: PF-06863135 1 mcg/kg IV | Part 1: PF-06863135 3 mcg/kg IV | Part 1: PF-06863135 10 mcg/kg IV | Part 1: PF-06863135 30 mcg/kg IV | Part 1: PF-06863135 50 mcg/kg IV | Part 1: PF-06863135 80 mcg/kg SC | Part 1: PF-06863135 130 mcg/kg SC | Part 1: PF-06863135 215 mcg/kg SC | Part 1: PF-06863135 360 mcg/kg SC | Part 1: PF-06863135 600 mcg/kg SC | Part 1: PF-06863135 1000 mcg/kg SC | Part 1.1: PF-06863135 Priming Cohort Q1W SC | Part 1.1: PF-06863135 Priming Cohort Q2W SC | Part 1C: PF-06863135 + Lenalidomide SC | Part 1D: PF-06863135 + Pomalidomide SC | Part 1: PF-06863135 Total IV | Part 1: PF-06863135 Total SC | Part 1.1: PF-06863135 Total SC
Number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 5 | 6 | 6 | 4 | 4 | 4 | 6 | 6 | 7 | 13 | 4 | 9 | 23 | 30 | 20
Months | 0.4 [0.3 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 0.7 [0.3 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 1.1 [0.7 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 1.7 [0.6 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 1.6 [0.6 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 1.6 [0.6 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 2.9 [0.8 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 1.0 [0.7 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 1.0 [0.7 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 19.1 [4.8 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 10.2 [0.7 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 32.9 [0.7 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 8.0 [0.7 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 7.6 [3.9 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 12.7 [0.5 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 18.1 [1.7 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 6.7 [0.9 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 1.4 [0.6 to 2.6] | 4.8 [1.1 to 14.4] | 12.2 [3.9 to 19.2]

15. Secondary Outcome: Part 1: Overall Survival (OS)
Description: OS was defined as the time from start date of study treatment to date of death due to any cause. OS for participants not known to had died were censored on the date of last known alive.
Time Frame: Time from start date of study treatment to date of death due to any cause or last-known-alive date, whichever occurred first (maximum up to 63.31 months)
Population: mITT analysis set included all participants who have received at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1: PF-06863135 0.1 mcg/kg IV | Part 1: PF-06863135 0.3 mcg/kg IV | Part 1: PF-06863135 1 mcg/kg IV | Part 1: PF-06863135 3 mcg/kg IV | Part 1: PF-06863135 10 mcg/kg IV | Part 1: PF-06863135 30 mcg/kg IV | Part 1: PF-06863135 50 mcg/kg IV | Part 1: PF-06863135 80 mcg/kg SC | Part 1: PF-06863135 130 mcg/kg SC | Part 1: PF-06863135 215 mcg/kg SC | Part 1: PF-06863135 360 mcg/kg SC | Part 1: PF-06863135 600 mcg/kg SC | Part 1: PF-06863135 1000 mcg/kg SC | Part 1.1: PF-06863135 Priming Cohort Q1W SC | Part 1.1: PF-06863135 Priming Cohort Q2W SC | Part 1C: PF-06863135 + Lenalidomide SC | Part 1D: PF-06863135 + Pomalidomide SC | Part 1: PF-06863135 Total IV | Part 1: PF-06863135 Total SC | Part 1.1: PF-06863135 Total SC
Number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 5 | 6 | 6 | 4 | 4 | 4 | 6 | 6 | 7 | 13 | 4 | 9 | 23 | 30 | 20
Months | 8.2 [4.4 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 8.4 [1.9 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 11.2 [4.4 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 8.1 [1.7 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 16.2 [9.4 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 14.8 [2.4 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 18.0 [5.0 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 1.7 [0.8 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | NA [3.8 to NA] — The median and upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 19.1 [8.8 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 14.0 [3.0 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 32.9 [12.0 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | NA [2.2 to NA] — The median and upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 8.3 [3.9 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | NA [1.1 to NA] — The median and upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 31.3 [28.3 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | NA [5.7 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 12.0 [7.9 to 17.1] | 17.3 [6.2 to 44.8] | NA [5.4 to NA] — The median and upper limit of 95% CI was not estimable due to insufficient number of participants with events.

16. Secondary Outcome: Part 1: Percentage of Participants With Negative Minimal Residual Disease (MRD) Using IMWG MRD Criteria
Description: MRD negativity rate: percentage of participants with negative MRD (assessed by central laboratory) per IMWG criteria at any time from date of first dose until first documentation of confirmed progression, death or start of new anticancer therapy, whichever occurred first. Progression was defined as appearance of local, regional, distant disease of same type after CR or progression of pre-existing lesions. It didn't include second primary malignancies of unrelated types. MRD negativity was defined by two thresholds, 10^-5 and 10^-6.
Time Frame: Anytime from date of first dose until the first documentation of confirmed PD, death or start of new anticancer therapy, whichever occurred first (maximum up to 63.31 months)
Population: Safety Analysis set included all participants who received at least 1 full or partial dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: PF-06863135 0.1 mcg/kg IV | Part 1: PF-06863135 0.3 mcg/kg IV | Part 1: PF-06863135 1 mcg/kg IV | Part 1: PF-06863135 3 mcg/kg IV | Part 1: PF-06863135 10 mcg/kg IV | Part 1: PF-06863135 30 mcg/kg IV | Part 1: PF-06863135 50 mcg/kg IV | Part 1: PF-06863135 80 mcg/kg SC | Part 1: PF-06863135 130 mcg/kg SC | Part 1: PF-06863135 215 mcg/kg SC | Part 1: PF-06863135 360 mcg/kg SC | Part 1: PF-06863135 600 mcg/kg SC | Part 1: PF-06863135 1000 mcg/kg SC | Part 1.1: PF-06863135 Priming Cohort Q1W SC | Part 1.1: PF-06863135 Priming Cohort Q2W SC | Part 1C: PF-06863135 + Lenalidomide SC | Part 1D: PF-06863135 + Pomalidomide SC | Part 1: PF-06863135 Total IV | Part 1: PF-06863135 Total SC | Part 1.1: PF-06863135 Total SC
Number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 5 | 6 | 6 | 4 | 4 | 4 | 6 | 6 | 7 | 13 | 4 | 9 | 23 | 30 | 20
Percentage of participants
  10^-5 threshold MRD | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 50.00 | 0 | 16.67 | 16.67 | 28.57 | 38.46 | 25.00 | 0 | 0 | 13.33 | 35.00
  10^-6 threshold MRD | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 25.00 | 0 | 16.67 | 16.67 | 0 | 30.77 | 0 | 0 | 0 | 10.00 | 20.00

17. Secondary Outcome: Part 1: Maximum Observed Concentration (Cmax) of PF-06863135
Description: Cmax of PF-06863135 was measured in this outcome measure. Total is free and bound drug in the body.
Time Frame: 0 hours (h) on Day 1 of Cycle (C) 0; 0, 2 and 4h on Day 1 of C1 and C2
Population: Pharmacokinetic (PK) parameter analysis set was defined as all enrolled participants treated who had sufficient information to estimate at least 1 of the PF- 06863135 PK parameters of interest. All participants reported under "Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. Here, "Number Analyzed" signifies number of participants evaluable at specified rows.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Part 1: PF-06863135 0.1 mcg/kg IV | Part 1: PF-06863135 0.3 mcg/kg IV | Part 1: PF-06863135 1 mcg/kg IV | Part 1: PF-06863135 3 mcg/kg IV | Part 1: PF-06863135 10 mcg/kg IV | Part 1: PF-06863135 30 mcg/kg IV | Part 1: PF-06863135 50 mcg/kg IV | Part 1: PF-06863135 80 mcg/kg SC | Part 1: PF-06863135 130 mcg/kg SC | Part 1: PF-06863135 215 mcg/kg SC | Part 1: PF-06863135 360 mcg/kg SC | Part 1: PF-06863135 600 mcg/kg SC | Part 1: PF-06863135 1000 mcg/kg SC | Part 1.1: PF-06863135 Priming Cohort Q1W SC | Part 1.1: PF-06863135 Priming Cohort Q2W SC | Part 1C: PF-06863135 + Lenalidomide SC | Part 1D: PF-06863135 + Pomalidomide SC
Number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 5 | 6 | 6 | 4 | 4 | 4 | 6 | 6 | 6 | 12 | 4 | 9
Micrograms per milliliter
  Total PF-06863135: Cycle 0 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 10 | 4 | 8
  Total PF-06863135: Cycle 0 Day 1 |  |  |  |  |  |  |  |  |  |  |  |  |  | 3.639 (21) | 4.216 (42) | 2.144 (96) | 2.277 (51)
  Total PF-06863135: Cycle 1 Day 1: number analyzed (Participants) | 2 | 2 | 2 | 3 | 2 | 5 | 6 | 6 | 4 | 4 | 4 | 6 | 6 | 6 | 11 | 4 | 9
  Total PF-06863135: Cycle 1 Day 1 | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 0.00168 and 0.00282. | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 0.00287 and 0.00439 | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 0.0122 and 0.0133. | 0.05363 (36) | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 0.164 and 0.297. | 0.6044 (27) | 0.8725 (41) | 0.2866 (46) | 0.9076 (24) | 1.220 (25) | 2.568 (42) | 3.802 (12) | 3.620 (53) | 9.927 (18) | 8.710 (54) | 5.513 (141) | 5.814 (36)
  Total PF-06863135: Cycle 2 Day 1: number analyzed (Participants) | 0 | 2 | 1 | 2 | 1 | 3 | 3 | 5 | 4 | 3 | 4 | 6 | 6 | 4 | 4 | 1 | 2
  Total PF-06863135: Cycle 2 Day 1 |  | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 0.475 and 0.624. | NA — Since only 1 participant evaluable, summary statistics could not be calculated. Individual participant data was 0.219. | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 0.151 and 0.233. | NA — Since only 1 participant evaluable, summary statistics could not be calculated. Individual participant data was 0.440. | 0.9924 (8) | 1.684 (23) | 0.6904 (55) | 2.108 (38) | 3.021 (24) | 5.748 (16) | 11.92 (28) | 12.98 (26) | 25.74 (19) | 12.03 (67) | NA — Since only 1 participant evaluable, summary statistics could not be calculated. Individual participant data was 16.6. | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 10.8 and 12.0.
  Free PF-06863135: Cycle 0 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 10 | 4 | 9
  Free PF-06863135: Cycle 0 Day 1 |  |  |  |  |  |  |  |  |  |  |  |  |  | 0.9445 (59) | 1.087 (79) | 0.5165 (83) | 0.8080 (59)
  Free PF-06863135: Cycle 1 Day 1: number analyzed (Participants) | 2 | 2 | 2 | 3 | 2 | 5 | 6 | 6 | 4 | 4 | 4 | 6 | 6 | 6 | 11 | 4 | 9
  Free PF-06863135: Cycle 1 Day 1 | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 0.000 and 0.000. | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 0.000 and 0.000. | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 0.000 and 0.000. | 0.0008828 (1.23) | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 0.0760 and 0.153. | 0.1851 (40) | 0.3015 (75) | 0.09913 (36) | 0.2479 (28) | 0.5916 (47) | 0.8304 (131) | 0.9875 (52) | 0.8266 (66) | 2.088 (106) | 2.485 (91) | 1.185 (90) | 2.150 (76)
  Free PF-06863135: Cycle 2 Day 1: number analyzed (Participants) | 0 | 2 | 1 | 2 | 1 | 3 | 3 | 5 | 4 | 3 | 4 | 6 | 6 | 4 | 4 | 1 | 2
  Free PF-06863135: Cycle 2 Day 1 |  | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 0.000 and 0.000. | NA — Since only 1 participant evaluable, summary statistics could not be calculated. Individual participant data was 0.000. | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 0.000 and 0.000. | NA (NA) — Since only 1 participant evaluable, summary statistics could not be calculated. Individual participant data was 0.103. | 0.2855 (37) | 0.2955 (4) | 0.1794 (40) | 0.3998 (41) | 1.473 (79) | 1.605 (182) | 7.981 (79) | 3.953 (156) | 11.00 (186) | 5.323 (69) | NA — Since only 1 participant evaluable, summary statistics could not be calculated. Individual participant data was 2.53. | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 9.65 and 12.1.

18. Secondary Outcome: Part 1: Area Under the Concentration-Time Profile From Time 0 to End of Dosing Interval (AUCtau)
Description: Area under the concentration curve from time 0 to end of dosing interval (AUCtau) was measured in this outcome measure. Total is free and bound drug in the body.
Time Frame: 0 hours (h) on Day 1 of Cycle (C) 0; 0, 2 and 4h on Day 1 of C1 and C2
Population: PK parameter analysis set was defined as all enrolled participants treated who had sufficient information to estimate at least 1 of the PF- 06863135 PK parameters of interest. All participants reported under "Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. Here, "Number Analyzed" signifies number of participants evaluable at specified rows.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram*day per milliliter
Arm/Group | Part 1: PF-06863135 0.1 mcg/kg IV | Part 1: PF-06863135 0.3 mcg/kg IV | Part 1: PF-06863135 1 mcg/kg IV | Part 1: PF-06863135 3 mcg/kg IV | Part 1: PF-06863135 10 mcg/kg IV | Part 1: PF-06863135 30 mcg/kg IV | Part 1: PF-06863135 50 mcg/kg IV | Part 1: PF-06863135 80 mcg/kg SC | Part 1: PF-06863135 130 mcg/kg SC | Part 1: PF-06863135 215 mcg/kg SC | Part 1: PF-06863135 360 mcg/kg SC | Part 1: PF-06863135 600 mcg/kg SC | Part 1: PF-06863135 1000 mcg/kg SC | Part 1.1: PF-06863135 Priming Cohort Q1W SC | Part 1.1: PF-06863135 Priming Cohort Q2W SC | Part 1C: PF-06863135 + Lenalidomide SC | Part 1D: PF-06863135 + Pomalidomide SC
Number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 5 | 6 | 6 | 4 | 4 | 4 | 6 | 6 | 6 | 12 | 4 | 9
Microgram*day per milliliter
  Total PF-06863135: Cycle 0 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 10 | 3 | 8
  Total PF-06863135: Cycle 0 Day 1 |  |  |  |  |  |  |  |  |  |  |  |  |  | 16.82 (20) | 16.93 (46) | 9.643 (148) | 10.91 (37)
  Total PF-06863135: Cycle 1 Day 1: number analyzed (Participants) | 1 | 2 | 2 | 3 | 2 | 5 | 5 | 3 | 3 | 2 | 4 | 6 | 4 | 5 | 8 | 3 | 6
  Total PF-06863135: Cycle 1 Day 1 | NA — Since only 1 participant evaluable, summary statistics could not be calculated. Individual participant data was 0.00829. | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 0.00933 and 0.0136. | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 0.0483 and 0.0484. | 0.1654 (74) | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 0.763 and 0.877. | 2.190 (11) | 3.322 (40) | 1.182 (58) | 4.426 (17) | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 4.35 and 6.09. | 12.58 (26) | 17.92 (29) | 25.53 (36) | 58.93 (14) | 93.96 (53) | 54.78 (16) | 31.92 (45)
  Total PF-06863135: Cycle 2 Day 1: number analyzed (Participants) | 0 | 1 | 1 | 0 | 0 | 2 | 2 | 2 | 4 | 0 | 2 | 6 | 4 | 3 | 4 | 0 | 2
  Total PF-06863135: Cycle 2 Day 1 |  | NA — Since only 1 participant evaluable, summary statistics could not be calculated. Individual participant data was 0.0276. | NA — Since only 1 participant evaluable, summary statistics could not be calculated. Individual participant data was 0.0790. |  |  | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 3.88 and 4.36. | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 7.91 and 8.10. | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 3.77 and 10.1. | 13.47 (39) |  | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 32.2 and 42.2. | 76.83 (30) | 88.92 (31) | 173.4 (21) | 148.1 (65) |  | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 71.7 and 77.8.
  Free PF-06863135: Cycle 0 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 10 | 3 | 8
  Free PF-06863135: Cycle 0 Day 1 |  |  |  |  |  |  |  |  |  |  |  |  |  | 4.111 (49) | 5.054 (73) | 2.447 (92) | 3.487 (50)
  Free PF-06863135: Cycle 1 Day 1: number analyzed (Participants) | 2 | 2 | 2 | 3 | 2 | 5 | 5 | 3 | 3 | 2 | 4 | 6 | 4 | 5 | 8 | 3 | 6
  Free PF-06863135: Cycle 1 Day 1 | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 0.000 and 0.000. | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 0.000 and 0.000. | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 0.000 and 0.000. | 0.0009462 (1.95) | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 0.261 and 0.618. | 0.7801 (24) | 1.206 (62) | 0.3344 (72) | 1.478 (23) | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 2.67 and 3.29. | 4.362 (103) | 4.909 (42) | 6.564 (33) | 11.92 (109) | 34.13 (60) | 8.896 (12) | 11.40 (91)
  Free PF-06863135: Cycle 2 Day 1: number analyzed (Participants) | 0 | 2 | 1 | 2 | 1 | 3 | 2 | 2 | 4 | 0 | 2 | 6 | 4 | 3 | 4 | 0 | 2
  Free PF-06863135: Cycle 2 Day 1 |  | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 0.000 and 0.000. | NA — Since only 1 participant evaluable, summary statistics could not be calculated. Individual participant data was 0.000. | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 0.000 and 0.000. | NA — Since only 1 participant evaluable, summary statistics could not be calculated. Individual participant data was 0.000. | 0.05280 (2.59) | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 1.51 and 1.57. | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 0.000 and 2.15. | 2.572 (49) |  | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 4.43 and 6.57. | 45.14 (113) | 34.18 (155) | 45.63 (128) | 66.20 (63) |  | NA (NA) — Since there were only 2 participants evaluable, summary statistics was not calculated. Individual participants data was 64.2 and 71.2.

19. Secondary Outcome: Part 1C and Part 1D: Plasma Concentration of Lenalidomide and Pomalidomide
Description: Plasma concentration of lenalidomide and pomalidomide was measured in this outcome measure.
Time Frame: Cycle 1 (0 hours post dose on Day 1, 8 and 15); Cycle 2 (0 hours on Day 15)
Population: PK Concentration Analysis Set was defined as all participants randomized and treated who had at least 1 measurable PF-06863135 concentration.
Measure: Median (Full Range); unit: nanogram/milliliter
Arm/Group | Part 1C: PF-06863135 + Lenalidomide SC | Part 1D: PF-06863135 + Pomalidomide SC
Number analyzed (Participants) | 4 | 9
nanogram/milliliter
  Cycle 1 Day 1 | NA [NA to NA] — Median, lower limit and upper limit was not estimable as the concentration was below the lower limit of quantification (LLOQ) of 1.00 nanogram per milliliter (ng/mL). | NA [NA to NA] — Median, lower limit and upper limit was not estimable as the concentration was below the lower limit of quantification (LLOQ) of 1.00 nanogram per milliliter (ng/mL).
  Cycle 1 Day 8 | 70.70 [70.7 to 70.7] | 13.60 [0.000 to 57.8]
  Cycle 1 Day 15 | 70.60 [70.6 to 70.6] | 32.70 [0.000 to 49.1]
  Cycle 2 Day 15 | 36.70 [20.2 to 234] | 0.0000 [0.000 to 7.41]

20. Secondary Outcome: Part 1: Number of Participants With Anti-Drug Antibodies (ADA) and Neutralizing Antibodies (NAb) Against PF-06863135
Description: Number of participants with ADA and NAb against PF-06863135 were reported in this outcome measure. A participant was ADA (or NAb) positive if: (1) baseline titer was missing or negative and participant had >= 1 post-treatment positive titer (treatment-induced), or (2) positive titer at baseline and had a >= 4-folder dilution increase in titer from baseline in >= 1 post-treatment sample (treatment-boosted).
Time Frame: From first dose of the study treatment (Day 1) up to end of study treatment (maximum up to 63.31 months)
Population: The immunogenicity analysis set was defined as participants who received at least 1 dose of study treatment and have at least 1 ADA sample collected. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: PF-06863135 0.1 mcg/kg IV | Part 1: PF-06863135 0.3 mcg/kg IV | Part 1: PF-06863135 1 mcg/kg IV | Part 1: PF-06863135 3 mcg/kg IV | Part 1: PF-06863135 10 mcg/kg IV | Part 1: PF-06863135 30 mcg/kg IV | Part 1: PF-06863135 50 mcg/kg IV | Part 1: PF-06863135 80 mcg/kg SC | Part 1: PF-06863135 130 mcg/kg SC | Part 1: PF-06863135 215 mcg/kg SC | Part 1: PF-06863135 360 mcg/kg SC | Part 1: PF-06863135 600 mcg/kg SC | Part 1: PF-06863135 1000 mcg/kg SC | Part 1.1: PF-06863135 Priming Cohort Q1W SC | Part 1.1: PF-06863135 Priming Cohort Q2W SC | Part 1C: PF-06863135 + Lenalidomide SC | Part 1D: PF-06863135 + Pomalidomide SC
Number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 5 | 6 | 6 | 4 | 4 | 4 | 6 | 6 | 6 | 13 | 4 | 9
Participants
  ADA positive | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  NAb positive | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: Part 1: Concentration of Soluble Cytokines in Serum
Description: The concentration of Interleukin-2, Interleukin-6, Interferon-gamma and tumor necrosis factor-alpha were measured in this outcome measure. Cycle = C.
Time Frame: Part 1: C1 (0, 2, 4 & 8 hours [h] post dose on Day [D] 1, 24h post dose on D2, 72h post dose on D3); Part 1.1, 1C & 1D: C0 (0, 2, 4 & 8h post dose on D1, 24h post dose on D2); C1 (0, 2, 4 & 8h post dose on D1, 24h post dose on D2, 72h post dose on D3)
Population: The Pharmacodynamic (PD)/Biomarker analysis set included all enrolled participants with at least 1 of the PD/Biomarkers evaluated at pre- and/or post-dose. Here, "Number Analyzed" signifies participants evaluable for specified rows.
Measure: Median (Full Range); unit: Picogram per milliliter
Arm/Group | Part 1: PF-06863135 0.1 mcg/kg IV | Part 1: PF-06863135 0.3 mcg/kg IV | Part 1: PF-06863135 1 mcg/kg IV | Part 1: PF-06863135 3 mcg/kg IV | Part 1: PF-06863135 10 mcg/kg IV | Part 1: PF-06863135 30 mcg/kg IV | Part 1: PF-06863135 50 mcg/kg IV | Part 1: PF-06863135 80 mcg/kg SC | Part 1: PF-06863135 130 mcg/kg SC | Part 1: PF-06863135 215 mcg/kg SC | Part 1: PF-06863135 360 mcg/kg SC | Part 1: PF-06863135 600 mcg/kg SC | Part 1: PF-06863135 1000 mcg/kg SC | Part 1.1: PF-06863135 Priming Cohort Q1W SC | Part 1.1: PF-06863135 Priming Cohort Q2W SC | Part 1C: PF-06863135 + Lenalidomide SC | Part 1D: PF-06863135 + Pomalidomide SC
Number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 5 | 6 | 6 | 4 | 4 | 4 | 6 | 6 | 7 | 13 | 4 | 9
Picogram per milliliter
  Interleukin-2: Cycle 0; 0 hours: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 13 | 4 | 8
  Interleukin-2: Cycle 0; 0 hours |  |  |  |  |  |  |  |  |  |  |  |  |  | 2.10 [2.1 to 2.1] | 2.10 [2.1 to 2.1] | 2.10 [2.1 to 2.1] | 2.10 [2.1 to 2.1]
  Interleukin-2: Cycle 0; 2 hours: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 13 | 4 | 8
  Interleukin-2: Cycle 0; 2 hours |  |  |  |  |  |  |  |  |  |  |  |  |  | 2.10 [2.1 to 9.1] | 2.10 [2.1 to 55.0] | 2.10 [2.1 to 2.1] | 2.10 [2.1 to 10.5]
  Interleukin-2: Cycle 0; 4 hours: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 13 | 4 | 8
  Interleukin-2: Cycle 0; 4 hours |  |  |  |  |  |  |  |  |  |  |  |  |  | 2.70 [2.1 to 19.7] | 3.60 [2.1 to 247.4] | 2.10 [2.1 to 6.5] | 2.40 [2.1 to 20.9]
  Interleukin-2: Cycle 0; 8 hours: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 13 | 4 | 8
  Interleukin-2: Cycle 0; 8 hours |  |  |  |  |  |  |  |  |  |  |  |  |  | 14.30 [2.1 to 487.8] | 17.90 [2.1 to 118.1] | 2.10 [2.1 to 82.0] | 2.10 [2.1 to 1063.8]
  Interleukin-2: Cycle 0; 24 hours: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 13 | 4 | 9
  Interleukin-2: Cycle 0; 24 hours |  |  |  |  |  |  |  |  |  |  |  |  |  | 2.10 [2.1 to 12.2] | 2.10 [2.1 to 15.5] | 2.10 [2.1 to 2.3] | 2.10 [2.1 to 7.1]
  Interleukin-2: Cycle 1; 0 hours: number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 5 | 6 | 6 | 4 | 4 | 4 | 6 | 6 | 6 | 12 | 4 | 9
  Interleukin-2: Cycle 1; 0 hours | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 24.0] | 5.00 [5.0 to 37.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [2.1 to 5.0] | 2.10 [2.1 to 2.1] | 2.10 [2.1 to 2.1] | 2.10 [2.1 to 2.1] | 2.10 [2.1 to 2.1] | 2.10 [2.1 to 2.1]
  Interleukin-2: Cycle 1; 2 hours: number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 4 | 4 | 6 | 4 | 4 | 4 | 6 | 6 | 6 | 12 | 4 | 8
  Interleukin-2: Cycle 1; 2 hours | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 12.50 [5.0 to 112.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [2.1 to 5.0] | 2.10 [2.1 to 2.1] | 2.10 [2.1 to 2.1] | 2.10 [2.1 to 2.1] | 2.10 [2.1 to 2.1] | 2.10 [2.1 to 2.1]
  Interleukin-2: Cycle 1; 4 hours: number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 4 | 5 | 6 | 4 | 4 | 4 | 6 | 6 | 6 | 12 | 4 | 9
  Interleukin-2: Cycle 1; 4 hours | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.50 [5.0 to 6.0] | 53.00 [5.0 to 80.0] | 83.00 [21.0 to 202.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 12.0] | 5.00 [5.0 to 5.0] | 5.50 [5.0 to 7.0] | 5.00 [2.1 to 6.7] | 2.10 [2.1 to 34.9] | 2.10 [2.1 to 2.2] | 2.10 [2.1 to 2.1] | 2.10 [2.1 to 2.1] | 2.10 [2.1 to 2.1]
  Interleukin-2: Cycle 1; 8 hours: number analyzed (Participants) | 2 | 3 | 2 | 2 | 2 | 4 | 5 | 6 | 4 | 4 | 4 | 6 | 6 | 6 | 11 | 4 | 9
  Interleukin-2: Cycle 1; 8 hours | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 11.0 [5.0 to 43.0] | 5.00 [5.0 to 52.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 50.0] | 8.50 [5.0 to 15.0] | 12.50 [5.0 to 39.0] | 5.00 [2.1 to 20.0] | 2.10 [2.1 to 55.7] | 2.10 [2.1 to 18.3] | 2.10 [2.1 to 2.1] | 2.10 [2.1 to 2.4] | 2.10 [2.1 to 2.1]
  Interleukin-2: Cycle 1; 24 hours: number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 5 | 5 | 6 | 4 | 4 | 4 | 6 | 6 | 6 | 12 | 4 | 9
  Interleukin-2: Cycle 1; 24 hours | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 9.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [2.1 to 5.0] | 2.10 [2.1 to 5.8] | 2.10 [2.1 to 2.7] | 2.10 [2.1 to 8.0] | 2.10 [2.1 to 7.4] | 2.10 [2.1 to 7.2]
  Interleukin-2: Cycle 1; 72 hours: number analyzed (Participants) | 2 | 3 | 2 | 3 | 1 | 5 | 5 | 6 | 4 | 4 | 4 | 6 | 6 | 6 | 12 | 4 | 8
  Interleukin-2: Cycle 1; 72 hours | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 14.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [2.1 to 5.0] | 2.10 [2.1 to 2.1] | 2.10 [2.1 to 2.1] | 2.10 [2.1 to 2.1] | 2.10 [2.1 to 4.7] | 2.10 [2.1 to 3.5]
  Interleukin-6: Cycle 0; 0 hours: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 13 | 4 | 8
  Interleukin-6: Cycle 0; 0 hours |  |  |  |  |  |  |  |  |  |  |  |  |  | 2.00 [2.0 to 4.9] | 2.00 [2.0 to 17.4] | 2.00 [2.0 to 2.9] | 2.00 [2.0 to 2.5]
  Interleukin-6: Cycle 0; 2 hours: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 13 | 4 | 8
  Interleukin-6: Cycle 0; 2 hours |  |  |  |  |  |  |  |  |  |  |  |  |  | 2.10 [2.0 to 10.8] | 2.00 [2.0 to 60.5] | 2.00 [2.0 to 3.6] | 2.00 [2.0 to 2.2]
  Interleukin-6: Cycle 0; 4 hours: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 13 | 4 | 8
  Interleukin-6: Cycle 0; 4 hours |  |  |  |  |  |  |  |  |  |  |  |  |  | 11.50 [3.2 to 63.6] | 10.40 [2.0 to 843.7] | 3.75 [2.0 to 17.1] | 5.25 [2.0 to 88.5]
  Interleukin-6: Cycle 0; 8 hours: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 13 | 4 | 7
  Interleukin-6: Cycle 0; 8 hours |  |  |  |  |  |  |  |  |  |  |  |  |  | 88.40 [14.8 to 1821.1] | 129.90 [2.0 to 1028.0] | 3.70 [2.2 to 670.4] | 2.00 [2.0 to 169.8]
  Interleukin-6: Cycle 0; 24 hours: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 13 | 4 | 9
  Interleukin-6: Cycle 0; 24 hours |  |  |  |  |  |  |  |  |  |  |  |  |  | 201.40 [15.1 to 428.4] | 122.70 [2.6 to 2396.8] | 8.50 [5.3 to 1651.0] | 33.60 [4.7 to 882.2]
  Interleukin-6: Cycle 1; 0 hours: number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 5 | 6 | 6 | 4 | 4 | 4 | 6 | 6 | 6 | 12 | 4 | 9
  Interleukin-6: Cycle 1; 0 hours | 7.00 [5.0 to 9.0] | 5.00 [5.0 to 5.0] | 6.50 [5.0 to 8.0] | 5.00 [5.0 to 12.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 32.0] | 5.00 [5.0 to 7.0] | 5.00 [5.0 to 32.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 6.50 [5.0 to 23.0] | 5.00 [2.0 to 5.0] | 2.00 [2.0 to 28.1] | 59.20 [9.6 to 370.9] | 24.50 [2.1 to 212.3] | 9.30 [2.0 to 219.5] | 2.00 [2.0 to 146.8]
  Interleukin-6: Cycle 1; 2 hours: number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 4 | 4 | 6 | 4 | 4 | 4 | 6 | 6 | 6 | 12 | 4 | 9
  Interleukin-6: Cycle 1; 2 hours | 6.00 [5.0 to 7.0] | 5.00 [5.0 to 5.0] | 17.00 [5.0 to 29.0] | 5.00 [5.0 to 14.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 29.0] | 9.50 [5.0 to 56.0] | 5.00 [5.0 to 43.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 6.50 [5.0 to 20.0] | 5.00 [2.0 to 5.0] | 2.00 [2.0 to 151.6] | 56.45 [7.7 to 205.1] | 20.60 [2.7 to 150.5] | 8.05 [2.0 to 278.8] | 2.30 [2.0 to 200.5]
  Interleukin-6: Cycle 1; 4 hours: number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 4 | 5 | 6 | 4 | 4 | 4 | 6 | 6 | 6 | 12 | 4 | 8
  Interleukin-6: Cycle 1; 4 hours | 6.50 [5.0 to 8.0] | 5.00 [5.0 to 5.0] | 7.00 [5.0 to 9.0] | 5.00 [5.0 to 16.0] | 5.00 [5.0 to 5.0] | 106.00 [5.0 to 206.0] | 73.00 [15.0 to 813.0] | 5.00 [5.0 to 54.0] | 5.00 [5.0 to 12.0] | 5.00 [5.0 to 7.0] | 15.50 [5.0 to 71.0] | 5.00 [3.5 to 21.7] | 8.95 [2.0 to 20.0] | 58.70 [5.5 to 303.8] | 22.95 [3.2 to 187.4] | 7.45 [2.0 to 292.6] | 2.25 [2.0 to 165.0]
  Interleukin-6: Cycle 1; 8 hours: number analyzed (Participants) | 2 | 3 | 2 | 2 | 2 | 4 | 5 | 6 | 4 | 4 | 4 | 6 | 6 | 5 | 11 | 4 | 9
  Interleukin-6: Cycle 1; 8 hours | 5.50 [5.0 to 6.0] | 5.00 [5.0 to 5.0] | 6.50 [5.0 to 8.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 40.00 [5.0 to 327.0] | 25.00 [5.0 to 263.0] | 5.00 [5.00 to 33.0] | 8.00 [5.0 to 54.0] | 46.50 [5.0 to 67.0] | 184.50 [12.0 to 342.0] | 12.00 [5.0 to 33.6] | 24.85 [2.0 to 2080.9] | 52.50 [6.9 to 125.1] | 35.00 [5.1 to 174.8] | 12.80 [2.0 to 634.1] | 2.00 [2.0 to 621.5]
  Interleukin-6: Cycle 1; 24 hours: number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 5 | 5 | 6 | 4 | 4 | 3 | 6 | 6 | 6 | 12 | 4 | 8
  Interleukin-6: Cycle 1; 24 hours | 7.00 [5.0 to 9.0] | 5.00 [5.0 to 5.0] | 8.00 [5.0 to 11.0] | 5.00 [5.0 to 163.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 45.0] | 6.00 [5.0 to 18.0] | 7.00 [5.0 to 64.0] | 9.00 [5.0 to 13.0] | 16.50 [6.0 to 51.0] | 29.00 [13.0 to 209.0] | 21.50 [5.0 to 976.8] | 31.25 [2.3 to 250.0] | 129.65 [10.5 to 631.3] | 38.35 [3.5 to 250.3] | 12.15 [2.0 to 577.6] | 2.90 [2.0 to 78.7]
  Interleukin-6: Cycle 1; 72 hours: number analyzed (Participants) | 2 | 3 | 2 | 3 | 1 | 5 | 5 | 5 | 4 | 4 | 4 | 6 | 5 | 6 | 12 | 4 | 8
  Interleukin-6: Cycle 1; 72 hours | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 8.50 [5.0 to 12.0] | 5.00 [5.0 to 56.0] | 5.00 [5.0 to 5.0] | 7.00 [5.0 to 37.0] | 5.00 [5.0 to 11.0] | 10.00 [5.0 to 13.0] | 6.00 [5.0 to 9.0] | 10.50 [5.0 to 74.0] | 11.0 [5.0 to 946.0] | 18.50 [5.0 to 224.2] | 7.20 [2.0 to 45.1] | 89.20 [11.1 to 161.3] | 30.45 [2.0 to 170.4] | 12.25 [2.0 to 188.3] | 32.75 [2.0 to 1239.3]
  Interferon-gamma: Cycle 0; 0 hours: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 13 | 4 | 8
  Interferon-gamma: Cycle 0; 0 hours |  |  |  |  |  |  |  |  |  |  |  |  |  | 4.20 [4.2 to 4.2] | 4.20 [4.2 to 4.2] | 4.20 [4.2 to 4.2] | 4.20 [4.2 to 4.2]
  Interferon-gamma: Cycle 0; 2 hours: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 13 | 4 | 8
  Interferon-gamma: Cycle 0; 2 hours |  |  |  |  |  |  |  |  |  |  |  |  |  | 4.20 [4.2 to 4.2] | 4.20 [4.2 to 4.2] | 4.20 [4.2 to 4.2] | 4.20 [4.2 to 4.2]
  Interferon-gamma: Cycle 0; 4 hours: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 13 | 4 | 8
  Interferon-gamma: Cycle 0; 4 hours |  |  |  |  |  |  |  |  |  |  |  |  |  | 4.20 [4.2 to 13.8] | 4.20 [2.2 to 18.3] | 4.20 [4.2 to 4.2] | 4.20 [4.2 to 12.8]
  Interferon-gamma: Cycle 0; 8 hours: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 13 | 4 | 8
  Interferon-gamma: Cycle 0; 8 hours |  |  |  |  |  |  |  |  |  |  |  |  |  | 10.30 [4.2 to 487.8] | 7.20 [4.2 to 34.6] | 4.20 [4.2 to 26.3] | 4.20 [4.2 to 106.1]
  Interferon-gamma: Cycle 0; 24 hours: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 13 | 4 | 9
  Interferon-gamma: Cycle 0; 24 hours |  |  |  |  |  |  |  |  |  |  |  |  |  | 5.00 [4.2 to 28.4] | 7.40 [4.2 to 17.4] | 4.20 [4.2 to 25.6] | 4.20 [4.2 to 23.1]
  Interferon-gamma: Cycle 1; 0 hours: number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 5 | 6 | 6 | 4 | 4 | 4 | 6 | 6 | 6 | 12 | 4 | 9
  Interferon-gamma: Cycle 1; 0 hours | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 7.0] | 5.00 [5.0 to 164.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [4.2 to 5.0] | 4.20 [4.2 to 4.2] | 4.20 [4.2 to 4.2] | 4.20 [4.2 to 4.2] | 4.20 [4.2 to 4.2] | 4.20 [4.2 to 5.9]
  Interferon-gamma: Cycle 1; 2 hours: number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 4 | 4 | 6 | 4 | 4 | 4 | 6 | 6 | 6 | 12 | 4 | 9
  Interferon-gamma: Cycle 1; 2 hours | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [4.2 to 5.0] | 4.20 [4.2 to 4.2] | 4.20 [4.2 to 4.2] | 4.20 [4.2 to 4.2] | 4.20 [4.2 to 4.9] | 4.20 [4.2 to 7.3]
  Interferon-gamma: Cycle 1; 4 hours: number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 4 | 5 | 6 | 4 | 4 | 4 | 6 | 6 | 6 | 12 | 4 | 8
  Interferon-gamma: Cycle 1; 4 hours | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 9.00 [5.0 to 13.0] | 10.00 [5.0 to 33.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [4.2 to 5.0] | 4.20 [4.2 to 19.0] | 4.20 [4.2 to 4.2] | 4.20 [4.2 to 4.2] | 4.20 [4.2 to 4.2] | 4.20 [4.2 to 5.2]
  Interferon-gamma: Cycle 1; 8 hours: number analyzed (Participants) | 2 | 3 | 2 | 2 | 2 | 4 | 5 | 6 | 4 | 4 | 4 | 6 | 6 | 6 | 11 | 4 | 9
  Interferon-gamma: Cycle 1; 8 hours | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 8.50 [5.0 to 39.0] | 5.00 [5.0 to 16.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.50 [5.0 to 8.0] | 5.50 [5.0 to 22.0] | 5.00 [4.2 to 6.0] | 4.20 [4.2 to 56.9] | 4.20 [4.2 to 5.5] | 4.20 [4.2 to 4.2] | 4.20 [4.2 to 4.2] | 4.20 [4.2 to 7.0]
  Interferon-gamma: Cycle 1; 24 hours: number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 5 | 5 | 6 | 4 | 4 | 4 | 6 | 6 | 6 | 12 | 4 | 9
  Interferon-gamma: Cycle 1; 24 hours | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 9.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 7.00 [5.0 to 12.0] | 5.00 [5.0 to 20.0] | 5.00 [5.0 to 12.1] | 4.20 [4.2 to 5.9] | 4.20 [4.2 to 4.2] | 4.20 [4.2 to 4.2] | 4.20 [4.2 to 4.2] | 4.20 [4.2 to 20.4]
  Interferon-gamma: Cycle 1; 72 hours: number analyzed (Participants) | 2 | 3 | 2 | 3 | 1 | 5 | 5 | 6 | 4 | 4 | 4 | 6 | 6 | 6 | 12 | 4 | 8
  Interferon-gamma: Cycle 1; 72 hours | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [4.2 to 5.0] | 4.20 [0.4 to 4.2] | 4.20 [4.2 to 4.2] | 4.20 [4.2 to 4.2] | 4.20 [4.2 to 4.2] | 4.20 [4.2 to 8.4]
  Tumor necrosis factor-alpha: Cycle 0; 0 hours: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 13 | 4 | 8
  Tumor necrosis factor-alpha: Cycle 0; 0 hours |  |  |  |  |  |  |  |  |  |  |  |  |  | 1.70 [1.7 to 1.7] | 1.70 [1.7 to 17.7] | 2.00 [1.7 to 2.3] | 1.70 [1.7 to 1.7]
  Tumor necrosis factor-alpha: Cycle 0; 2 hours: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 13 | 4 | 8
  Tumor necrosis factor-alpha: Cycle 0; 2 hours |  |  |  |  |  |  |  |  |  |  |  |  |  | 1.70 [1.7 to 2.8] | 1.70 [1.7 to 75.6] | 1.70 [1.7 to 3.5] | 2.35 [1.7 to 6.2]
  Tumor necrosis factor-alpha: Cycle 0; 4 hours: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 13 | 4 | 8
  Tumor necrosis factor-alpha: Cycle 0; 4 hours |  |  |  |  |  |  |  |  |  |  |  |  |  | 3.30 [1.7 to 27.7] | 2.50 [1.7 to 164.2] | 2.60 [1.7 to 9.7] | 1.70 [1.7 to 8.9]
  Tumor necrosis factor-alpha: Cycle 0; 8 hours: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 13 | 4 | 8
  Tumor necrosis factor-alpha: Cycle 0; 8 hours |  |  |  |  |  |  |  |  |  |  |  |  |  | 9.70 [1.7 to 46.2] | 7.40 [1.7 to 39.2] | 3.05 [1.7 to 39.1] | 1.75 [1.7 to 114.2]
  Tumor necrosis factor-alpha: Cycle 0; 24 hours: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 13 | 4 | 9
  Tumor necrosis factor-alpha: Cycle 0; 24 hours |  |  |  |  |  |  |  |  |  |  |  |  |  | 3.80 [1.7 to 9.1] | 3.80 [1.7 to 15.1] | 3.15 [1.7 to 4.2] | 2.30 [1.7 to 8.5]
  Tumor necrosis factor-alpha: Cycle 1; 0 hours: number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 5 | 6 | 6 | 4 | 4 | 4 | 6 | 6 | 6 | 12 | 4 | 9
  Tumor necrosis factor-alpha: Cycle 1; 0 hours | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 41.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 25.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 37.0] | 5.00 [1.7 to 16.0] | 1.70 [1.7 to 18.4] | 1.70 [1.7 to 2.2] | 1.70 [1.7 to 10.3] | 3.15 [1.7 to 4.6] | 1.70 [1.7 to 3.3]
  Tumor necrosis factor-alpha: Cycle 1; 2 hours: number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 4 | 4 | 6 | 4 | 4 | 4 | 6 | 6 | 6 | 12 | 4 | 9
  Tumor necrosis factor-alpha: Cycle 1; 2 hours | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 8.0] | 8.50 [5.0 to 21.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [1.7 to 15.0] | 1.70 [1.7 to 25.5] | 1.70 [1.7 to 1.7] | 1.80 [1.7 to 14.7] | 2.55 [1.7 to 4.1] | 1.70 [1.7 to 6.5]
  Tumor necrosis factor-alpha: Cycle 1; 4 hours: number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 4 | 5 | 6 | 4 | 4 | 4 | 6 | 6 | 6 | 12 | 4 | 8
  Tumor necrosis factor-alpha: Cycle 1; 4 hours | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 11.0 [5.0 to 70.0] | 8.00 [5.0 to 138.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [1.7 to 12.0] | 1.70 [1.7 to 147.3] | 1.70 [1.7 to 2.7] | 1.70 [1.7 to 6.3] | 2.80 [1.7 to 4.0] | 1.70 [1.7 to 4.0]
  Tumor necrosis factor-alpha: Cycle 1; 8 hours: number analyzed (Participants) | 2 | 3 | 2 | 2 | 2 | 4 | 6 | 6 | 4 | 4 | 4 | 6 | 6 | 6 | 11 | 4 | 9
  Tumor necrosis factor-alpha: Cycle 1; 8 hours | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 6.0] | 5.00 [5.0 to 12.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 6.0] | 6.50 [5.0 to 35.0] | 8.00 [5.0 to 11.0] | 5.00 [1.7 to 27.0] | 1.70 [1.7 to 458.0] | 1.70 [1.7 to 1.9] | 1.70 [1.7 to 11.6] | 1.70 [1.7 to 5.3] | 1.70 [1.4 to 5.8]
  Tumor necrosis factor-alpha: Cycle 1; 24 hours: number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 5 | 5 | 6 | 4 | 4 | 4 | 6 | 6 | 6 | 12 | 4 | 9
  Tumor necrosis factor-alpha: Cycle 1; 24 hours | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 7.0] | 5.00 [5.0 to 12.0] | 5.00 [1.7 to 9.0] | 1.70 [1.7 to 2.0] | 1.70 [1.7 to 2.1] | 2.45 [1.7 to 8.0] | 2.90 [1.7 to 4.1] | 1.70 [1.7 to 6.2]
  Tumor necrosis factor-alpha: Cycle 1; 72 hours: number analyzed (Participants) | 2 | 3 | 2 | 3 | 1 | 5 | 5 | 6 | 4 | 4 | 4 | 6 | 6 | 6 | 12 | 4 | 8
  Tumor necrosis factor-alpha: Cycle 1; 72 hours | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 15.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 5.0] | 5.00 [5.0 to 10.0] | 5.00 [5.0 to 5.0] | 5.00 [1.7 to 5.0] | 1.70 [1.7 to 3.4] | 1.70 [1.7 to 4.2] | 1.70 [1.7 to 6.7] | 3.85 [1.7 to 6.9] | 1.70 [1.7 to 3.6]

22. Secondary Outcome: Part 2: Number of Participants With AEs, Serious AEs, Treatment Related AEs, Grade 3 or 4 AEs and Grade 5 AEs as Graded by NCI CTCAE v4.03
Description: as for outcome 4
Time Frame: From first dose of the study treatment (Day 1) up to 30 days after the last dose of study treatment (maximum up to of 32.3 months)
Population: Safety analysis set included all participants who received at least 1 full or partial dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: PF-06863135 SC
Number analyzed (Participants) | 15
Participants
  Participants with TEAEs | 15
  Participants with serious AEs | 12
  Participants with treatment related AEs | 13
  Participants with grade 3 or 4 AEs | 11
  Participants with grade 5 AEs | 3

23. Secondary Outcome: Part 2: Number of Participants With Shifts From Grade <=2 at Baseline to Grade 3 or 4 Post-Baseline in Hematology Parameters
Description: as for outcome 5
Time Frame: as for outcome 22
Population: Safety analysis set included all participants who received at least 1 full or partial dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: PF-06863135 SC
Number analyzed (Participants) | 15
Participants | 15

24. Secondary Outcome: Part 2: Number of Participants With Shifts From Grade <= 2 at Baseline to Grade 3 or 4 Post-Baseline in Clinical Chemistry Parameters
Description: as for outcome 6
Time Frame: as for outcome 22
Population: Safety analysis set included all participants who received at least 1 full or partial dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: PF-06863135 SC
Number analyzed (Participants) | 15
Participants | 8

25. Secondary Outcome: Part 2: Number of Participants With Shifts From Grade <=2 to Grade 3 or 4 Post-Baseline in Urinalysis
Description: as for outcome 7
Time Frame: as for outcome 22
Population: Safety analysis set included all participants who received at least 1 full or partial dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: PF-06863135 SC
Number analyzed (Participants) | 15
Participants | 0

26. Secondary Outcome: Part 2: CRR as Per IMWG Criteria
Description: as for outcome 10
Time Frame: From the first dose of study treatment until the first documented sCR or CR or new anti-cancer therapies or death, whichever occurred first (maximum up to 34.3 months)
Population: mITT analysis set included all participants who have received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 2A: PF-06863135 SC
Number analyzed (Participants) | 15
Percentage of participants | 33.3 [15.2 to 58.3]

27. Secondary Outcome: Part 2: DoCR as Per IMWG Criteria
Description: DoCR was defined for participants with confirmed complete response (sCR or CR) as the time from the first documentation of complete response to the first documentation of objective tumor progression or to death due to any cause, whichever occured first. sCR: complete response plus normal FLC ratio and absence of clonal cells in bone marrow biopsy by immunohistochemistry; CR: Negative immunofixation on serum and urine and disappearance of any soft tissue plasmacytomas and <5% plasma cells in bone marrow aspirates. Progression was defined as appearance of local, regional or distant disease of same type after CR or progression of pre-existing lesions. It didn't include second primary malignancies of unrelated types.
Time Frame: From the first documentation of complete response to the first documentation of tumor progression or death, whichever occurred first (maximum up to 34.3 months)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Months
Arm/Group | Part 2A: PF-06863135 SC
Number analyzed (Participants) | 5
Months | 9.4 [6.5 to NA] — Upper limit of 95% CI was not estimable due to insufficient number of participants with event.

28. Secondary Outcome: Part 2: TTR as Per IMWG Criteria
Description: as for outcome 9
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Median (Full Range); unit: Days
Arm/Group | Part 2A: PF-06863135 SC
Number analyzed (Participants) | 9
Days | 40.0 [8 to 262]

29. Secondary Outcome: Part 2: DOSD as Per IMWG Criteria
Description: as for outcome 13
Time Frame: Time from the first documentation of objective stable disease to the first documentation of objective tumor progression or to death due to any cause, whichever occurred first (maximum up to 34.3 months)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2A: PF-06863135 SC
Number analyzed (Participants) | 12
Months | 11.6 [1.9 to NA] — Upper limit of 95% CI was not estimable due to insufficient number of participants with event.

30. Secondary Outcome: Part 2: PFS as Per IMWG Criteria
Description: as for outcome 14
Time Frame: From start date of study treatment to date of first documentation of progression or death due to any cause, whichever occurred first (maximum up to 34.3 months)
Population: mITT analysis set included all participants who have received at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2A: PF-06863135 SC
Number analyzed (Participants) | 15
Months | 10.4 [1.2 to 20.0]

31. Secondary Outcome: Part 2: OS
Description: as for outcome 15
Time Frame: Time from start date of study treatment to date of death due to any cause or last-known-alive date, whichever occurred first (maximum up to 34.3 months)
Population: mITT analysis set included all participants who have received at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2A: PF-06863135 SC
Number analyzed (Participants) | 15
Months | 12.1 [4.2 to NA] — Upper limit of 95% CI was not estimable due to insufficient number of participants with events.

32. Secondary Outcome: Part 2: Percentage of Participants With Negative MRD After Treatment With PF-06863135 Using IMWG MRD Criteria
Description: as for outcome 16
Time Frame: Anytime from date of first dose until the first documentation of confirmed PD, death or start of new anticancer therapy whichever occurred first (maximum up to 34.3 months)
Population: Safety Analysis set included all participants who received at least 1 full or partial dose of study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 2A: PF-06863135 SC
Number analyzed (Participants) | 15
Percentage of Participants
  10^-5 threshold MRD | 33.33
  10^-6 threshold MRD | 13.33

33. Secondary Outcome: Part 2: Number of Participants With ADA and NAb Against PF-06863135
Description: as for outcome 20
Time Frame: From first dose of the study treatment (Day 1) up to end of study treatment (maximum up to 34.3 months)
Population: The immunogenicity analysis set was defined as participants who received at least 1 dose of study treatment and have at least 1 ADA sample collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: PF-06863135 SC
Number analyzed (Participants) | 15
Participants
  ADA positive | 0
  NAb positive | 0

34. Secondary Outcome: Part 2: Concentration of Soluble Cytokines in Serum
Description: The concentration of Interleukin-2, Interleukin-6, Interferon-gamma and tumor necrosis factor-alpha were measured in this outcome measure.
Time Frame: Cycle 0 (0, 2, 4 and 8 hours post dose on Day 1, 24 hours post dose on Day 2); Cycle 1 (0, 2, 4 and 8 hours post dose on Day 1, 24 hours post dose on Day 2, 72 hours post dose on Day 3)
Population: The PD/Biomarker analysis set included all enrolled participants with at least 1 of the PD/Biomarkers evaluated at pre- and/or post-dose. All participants reported under "Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. Here, "Number Analyzed" signifies participants evaluable for specified rows.
Measure: Median (Full Range); unit: Picogram per milliliter
Arm/Group | Part 2A: PF-06863135 SC
Number analyzed (Participants) | 15
Picogram per milliliter
  Interleukin-2: Cycle 0; 0 hours: number analyzed (Participants) | 13
  Interleukin-2: Cycle 0; 0 hours | 2.10 [2.1 to 2.1]
  Interleukin-2: Cycle 0; 2 hours: number analyzed (Participants) | 13
  Interleukin-2: Cycle 0; 2 hours | 2.10 [2.1 to 27.5]
  Interleukin-2: Cycle 0; 4 hours: number analyzed (Participants) | 13
  Interleukin-2: Cycle 0; 4 hours | 2.10 [2.1 to 48.6]
  Interleukin-2: Cycle 0; 8 hours: number analyzed (Participants) | 13
  Interleukin-2: Cycle 0; 8 hours | 2.10 [2.1 to 10.6]
  Interleukin-2: Cycle 0; 24 hours: number analyzed (Participants) | 12
  Interleukin-2: Cycle 0; 24 hours | 2.10 [2.1 to 30.1]
  Interleukin-2: Cycle 1; 0 hours: number analyzed (Participants) | 14
  Interleukin-2: Cycle 1; 0 hours | 2.10 [2.1 to 2.1]
  Interleukin-2: Cycle 1; 2 hours: number analyzed (Participants) | 14
  Interleukin-2: Cycle 1; 2 hours | 2.10 [2.1 to 2.1]
  Interleukin-2: Cycle 1; 4 hours: number analyzed (Participants) | 14
  Interleukin-2: Cycle 1; 4 hours | 2.10 [2.1 to 2.1]
  Interleukin-2: Cycle 1; 8 hours: number analyzed (Participants) | 13
  Interleukin-2: Cycle 1; 8 hours | 2.10 [2.1 to 3.0]
  Interleukin-2: Cycle 1; 24 hours: number analyzed (Participants) | 13
  Interleukin-2: Cycle 1; 24 hours | 2.10 [2.1 to 2.1]
  Interleukin-2: Cycle 1; 72 hours: number analyzed (Participants) | 13
  Interleukin-2: Cycle 1; 72 hours | 2.10 [2.1 to 2.1]
  Interleukin-6: Cycle 0; 0 hours: number analyzed (Participants) | 13
  Interleukin-6: Cycle 0; 0 hours | 2.00 [2.0 to 63.1]
  Interleukin-6: Cycle 0; 2 hours: number analyzed (Participants) | 13
  Interleukin-6: Cycle 0; 2 hours | 2.00 [2.0 to 7.0]
  Interleukin-6: Cycle 0; 4 hours: number analyzed (Participants) | 13
  Interleukin-6: Cycle 0; 4 hours | 2.00 [2.0 to 23.1]
  Interleukin-6: Cycle 0; 8 hours: number analyzed (Participants) | 13
  Interleukin-6: Cycle 0; 8 hours | 2.00 [2.0 to 9.3]
  Interleukin-6: Cycle 0; 24 hours: number analyzed (Participants) | 12
  Interleukin-6: Cycle 0; 24 hours | 10.30 [2.0 to 2480.3]
  Interleukin-6: Cycle 1; 0 hours: number analyzed (Participants) | 14
  Interleukin-6: Cycle 1; 0 hours | 5.05 [2.0 to 156.0]
  Interleukin-6: Cycle 1; 2 hours: number analyzed (Participants) | 14
  Interleukin-6: Cycle 1; 2 hours | 2.00 [2.0 to 88.6]
  Interleukin-6: Cycle 1; 4 hours: number analyzed (Participants) | 14
  Interleukin-6: Cycle 1; 4 hours | 2.30 [2.0 to 78.9]
  Interleukin-6: Cycle 1; 8 hours: number analyzed (Participants) | 13
  Interleukin-6: Cycle 1; 8 hours | 2.00 [2.0 to 53.3]
  Interleukin-6: Cycle 1; 24 hours: number analyzed (Participants) | 13
  Interleukin-6: Cycle 1; 24 hours | 3.70 [2.0 to 466.7]
  Interleukin-6: Cycle 1; 72 hours: number analyzed (Participants) | 13
  Interleukin-6: Cycle 1; 72 hours | 7.50 [2.0 to 1231.3]
  Interferon-gamma: Cycle 0; 0 hours: number analyzed (Participants) | 13
  Interferon-gamma: Cycle 0; 0 hours | 4.20 [4.2 to 4.2]
  Interferon-gamma: Cycle 0; 2 hours: number analyzed (Participants) | 13
  Interferon-gamma: Cycle 0; 2 hours | 4.20 [4.2 to 4.2]
  Interferon-gamma: Cycle 0; 4 hours: number analyzed (Participants) | 13
  Interferon-gamma: Cycle 0; 4 hours | 4.20 [4.2 to 4.2]
  Interferon-gamma: Cycle 0; 8 hours: number analyzed (Participants) | 13
  Interferon-gamma: Cycle 0; 8 hours | 4.20 [3.0 to 4.2]
  Interferon-gamma: Cycle 0; 24 hours: number analyzed (Participants) | 12
  Interferon-gamma: Cycle 0; 24 hours | 4.20 [4.2 to 47.3]
  Interferon-gamma: Cycle 1; 0 hours: number analyzed (Participants) | 14
  Interferon-gamma: Cycle 1; 0 hours | 4.20 [4.2 to 4.2]
  Interferon-gamma: Cycle 1; 2 hours: number analyzed (Participants) | 14
  Interferon-gamma: Cycle 1; 2 hours | 4.20 [4.2 to 4.2]
  Interferon-gamma: Cycle 1; 4 hours: number analyzed (Participants) | 14
  Interferon-gamma: Cycle 1; 4 hours | 4.20 [2.2 to 4.2]
  Interferon-gamma: Cycle 1; 8 hours: number analyzed (Participants) | 13
  Interferon-gamma: Cycle 1; 8 hours | 4.20 [4.2 to 4.2]
  Interferon-gamma: Cycle 1; 24 hours: number analyzed (Participants) | 13
  Interferon-gamma: Cycle 1; 24 hours | 4.20 [4.2 to 7.5]
  Interferon-gamma: Cycle 1; 72 hours: number analyzed (Participants) | 13
  Interferon-gamma: Cycle 1; 72 hours | 4.20 [4.2 to 4.2]
  Tumor necrosis factor-alpha: Cycle 0; 0 hours: number analyzed (Participants) | 13
  Tumor necrosis factor-alpha: Cycle 0; 0 hours | 1.70 [1.7 to 2.8]
  Tumor necrosis factor-alpha: Cycle 0; 2 hours: number analyzed (Participants) | 13
  Tumor necrosis factor-alpha: Cycle 0; 2 hours | 1.70 [1.7 to 58.5]
  Tumor necrosis factor-alpha: Cycle 0; 4 hours: number analyzed (Participants) | 13
  Tumor necrosis factor-alpha: Cycle 0; 4 hours | 1.70 [1.7 to 20.8]
  Tumor necrosis factor-alpha: Cycle 0; 8 hours: number analyzed (Participants) | 13
  Tumor necrosis factor-alpha: Cycle 0; 8 hours | 1.70 [1.7 to 3.9]
  Tumor necrosis factor-alpha: Cycle 0; 24 hours: number analyzed (Participants) | 12
  Tumor necrosis factor-alpha: Cycle 0; 24 hours | 2.55 [1.7 to 12.7]
  Tumor necrosis factor-alpha: Cycle 1; 0 hours: number analyzed (Participants) | 14
  Tumor necrosis factor-alpha: Cycle 1; 0 hours | 1.70 [1.7 to 4.9]
  Tumor necrosis factor-alpha: Cycle 1; 2 hours: number analyzed (Participants) | 14
  Tumor necrosis factor-alpha: Cycle 1; 2 hours | 1.70 [1.7 to 5.2]
  Tumor necrosis factor-alpha: Cycle 1; 4 hours: number analyzed (Participants) | 14
  Tumor necrosis factor-alpha: Cycle 1; 4 hours | 1.70 [1.7 to 5.8]
  Tumor necrosis factor-alpha: Cycle 1; 8 hours: number analyzed (Participants) | 13
  Tumor necrosis factor-alpha: Cycle 1; 8 hours | 1.70 [1.7 to 3.6]
  Tumor necrosis factor-alpha: Cycle 1; 24 hours: number analyzed (Participants) | 13
  Tumor necrosis factor-alpha: Cycle 1; 24 hours | 1.70 [1.7 to 5.2]
  Tumor necrosis factor-alpha: Cycle 1; 72 hours: number analyzed (Participants) | 13
  Tumor necrosis factor-alpha: Cycle 1; 72 hours | 1.70 [1.7 to 2.9]

ADVERSE EVENTS:
Time Frame: Adverse events for Part 1: up to 43.3 months and for Part 2: up to 32.3 months; all-cause mortality for Part 1: 63.31 months and for Part 2: 34.3 months
Description: Same event may appear as both non-SAE and SAE but are distinct events. An event may be categorized as serious in 1 participant and non-serious in another, or a participant may have experienced both SAE and non-SAE. Safety analysis set included all participants who received at least 1 full or partial dose of study medication.
Arm/Group | Part 1: PF-06863135 0.1 mcg/kg IV | Part 1: PF-06863135 0.3 mcg/kg IV | Part 1: PF-06863135 1 mcg/kg IV | Part 1: PF-06863135 3 mcg/kg IV | Part 1: PF-06863135 10 mcg/kg IV | Part 1: PF-06863135 30 mcg/kg IV | Part 1: PF-06863135 50 mcg/kg IV | Part 1: PF-06863135 80 mcg/kg SC | Part 1: PF-06863135 130 mcg/kg SC | Part 1: PF-06863135 215 mcg/kg SC | Part 1: PF-06863135 360 mcg/kg SC | Part 1: PF-06863135 600 mcg/kg SC | Part 1: PF-06863135 1000 mcg/kg SC | Part 1.1: PF-06863135 Priming Cohort Q1W SC | Part 1.1: PF-06863135 Priming Cohort Q2W SC | Part 1C: PF-06863135 + Lenalidomide SC | Part 1D: PF-06863135 + Pomalidomide SC | Part 2A: PF-06863135 SC | Part 1: PF-06863135 Total IV | Part 1: PF-06863135 Total SC | Part 1.1: PF-06863135 Total SC
All-Cause Mortality (participants affected / at risk) | 2/2 | 2/3 | 2/2 | 3/3 | 2/2 | 4/5 | 4/6 | 5/6 | 1/4 | 3/4 | 3/4 | 3/6 | 2/6 | 3/7 | 4/13 | 2/4 | 4/9 | 10/15 | 19/23 | 17/30 | 7/20
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/3 | 0/2 | 3/3 | 0/2 | 2/5 | 5/6 | 4/6 | 1/4 | 3/4 | 3/4 | 4/6 | 5/6 | 6/7 | 9/13 | 2/4 | 8/9 | 12/15 | 11/23 | 20/30 | 15/20
Other Adverse Events (participants affected / at risk) | 2/2 | 3/3 | 2/2 | 3/3 | 2/2 | 5/5 | 6/6 | 6/6 | 4/4 | 4/4 | 4/4 | 6/6 | 6/6 | 7/7 | 13/13 | 4/4 | 9/9 | 13/15 | 23/23 | 30/30 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: PF-06863135 0.1 mcg/kg IV (N=2) | Part 1: PF-06863135 0.3 mcg/kg IV (N=3) | Part 1: PF-06863135 1 mcg/kg IV (N=2) | Part 1: PF-06863135 3 mcg/kg IV (N=3) | Part 1: PF-06863135 10 mcg/kg IV (N=2) | Part 1: PF-06863135 30 mcg/kg IV (N=5) | Part 1: PF-06863135 50 mcg/kg IV (N=6) | Part 1: PF-06863135 80 mcg/kg SC (N=6) | Part 1: PF-06863135 130 mcg/kg SC (N=4) | Part 1: PF-06863135 215 mcg/kg SC (N=4) | Part 1: PF-06863135 360 mcg/kg SC (N=4) | Part 1: PF-06863135 600 mcg/kg SC (N=6) | Part 1: PF-06863135 1000 mcg/kg SC (N=6) | Part 1.1: PF-06863135 Priming Cohort Q1W SC (N=7) | Part 1.1: PF-06863135 Priming Cohort Q2W SC (N=13) | Part 1C: PF-06863135 + Lenalidomide SC (N=4) | Part 1D: PF-06863135 + Pomalidomide SC (N=9) | Part 2A: PF-06863135 SC (N=15) | Part 1: PF-06863135 Total IV (N=23) | Part 1: PF-06863135 Total SC (N=30) | Part 1.1: PF-06863135 Total SC (N=20)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Extraocular muscle disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 2 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 3 | 1
Sudden death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 0 | 2 | 2 | 2 | 1 | 5 | 7 | 3 | 4 | 4
Adenovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Cytomegalovirus chorioretinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Encephalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Extradural abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes simplex oesophagitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 2 | 2
Salmonellosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Viral sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Immune effector cell-associated neurotoxicity syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neurotoxicity (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 2 | 1
Assisted suicide (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: PF-06863135 0.1 mcg/kg IV (N=2) | Part 1: PF-06863135 0.3 mcg/kg IV (N=3) | Part 1: PF-06863135 1 mcg/kg IV (N=2) | Part 1: PF-06863135 3 mcg/kg IV (N=3) | Part 1: PF-06863135 10 mcg/kg IV (N=2) | Part 1: PF-06863135 30 mcg/kg IV (N=5) | Part 1: PF-06863135 50 mcg/kg IV (N=6) | Part 1: PF-06863135 80 mcg/kg SC (N=6) | Part 1: PF-06863135 130 mcg/kg SC (N=4) | Part 1: PF-06863135 215 mcg/kg SC (N=4) | Part 1: PF-06863135 360 mcg/kg SC (N=4) | Part 1: PF-06863135 600 mcg/kg SC (N=6) | Part 1: PF-06863135 1000 mcg/kg SC (N=6) | Part 1.1: PF-06863135 Priming Cohort Q1W SC (N=7) | Part 1.1: PF-06863135 Priming Cohort Q2W SC (N=13) | Part 1C: PF-06863135 + Lenalidomide SC (N=4) | Part 1D: PF-06863135 + Pomalidomide SC (N=9) | Part 2A: PF-06863135 SC (N=15) | Part 1: PF-06863135 Total IV (N=23) | Part 1: PF-06863135 Total SC (N=30) | Part 1.1: PF-06863135 Total SC (N=20)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 1 | 1 | 2 | 4 | 3 | 4 | 3 | 3 | 4 | 3 | 5 | 6 | 9 | 1 | 3 | 6 | 14 | 22 | 15
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 3 | 0 | 2 | 3 | 1 | 3 | 3 | 2 | 4 | 2 | 4 | 2 | 7 | 12 | 6
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 1 | 2 | 3 | 4 | 3 | 4 | 4 | 5 | 6 | 3 | 4 | 3 | 3 | 3 | 9 | 26 | 7
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1 | 0 | 2 | 2 | 0 | 2 | 3 | 1 | 5 | 5 | 6 | 11 | 3 | 7 | 10 | 7 | 16 | 17
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 2 | 1 | 0 | 4 | 5 | 2 | 3 | 1 | 4 | 2 | 3 | 10 | 1 | 3 | 5 | 10 | 17 | 13
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 2 | 0 | 3 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 3 | 4 | 5 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 2 | 1 | 3 | 3 | 2 | 8 | 2 | 6 | 2 | 5 | 9 | 10
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 1 | 1 | 4 | 2 | 2 | 3 | 2 | 4 | 5 | 3 | 11 | 5
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 3 | 0 | 3 | 1 | 3 | 4 | 0 | 3 | 2 | 3 | 8 | 7
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 3 | 1 | 3 | 0 | 2 | 3 | 4
Fatigue (General disorders) | 0 | 0 | 1 | 1 | 0 | 4 | 1 | 1 | 1 | 0 | 1 | 2 | 2 | 3 | 8 | 1 | 7 | 7 | 7 | 7 | 11
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 5 | 5 | 6 | 6 | 4 | 6 | 6 | 0 | 16 | 12
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 2 | 1 | 4 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 1 | 2 | 1 | 1 | 1 | 0 | 6 | 3
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 2 | 1 | 3 | 2 | 5 | 2 | 0 | 7 | 4
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 4 | 5 | 2 | 2 | 2 | 2 | 6 | 4 | 6 | 11 | 1 | 3 | 3 | 10 | 18 | 17
Hypogammaglobulinaemia (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 4 | 1 | 1 | 0 | 0 | 3 | 4
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 0 | 3 | 0 | 1 | 3
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 2 | 1 | 1 | 1 | 1 | 4 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 1 | 3 | 5 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 2 | 0 | 5 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 3 | 1 | 2 | 3 | 3 | 1 | 6
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 3 | 3 | 1 | 5 | 0 | 1 | 1 | 1 | 10 | 6
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 0 | 4 | 2 | 1 | 5 | 0 | 1 | 3 | 4 | 10 | 6
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 2 | 0 | 0 | 3 | 1 | 3 | 4
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 2 | 3
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 6 | 2
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 3 | 2 | 2 | 0 | 0 | 4 | 4
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 1 | 3 | 0 | 2 | 6 | 1 | 5 | 4
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 1 | 1 | 1 | 2 | 1 | 2 | 5 | 3 | 1 | 7 | 5 | 7 | 7
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 3 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 3 | 0 | 0 | 1 | 0 | 5 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 1 | 1 | 4 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 4 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 3 | 0 | 1 | 2 | 2 | 5 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 5 | 0 | 2 | 2 | 0 | 1 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 3 | 3 | 2 | 5 | 3 | 2 | 6 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 2 | 7 | 1 | 3 | 3 | 2 | 7 | 9
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 4 | 0 | 1 | 1 | 1 | 4 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 2 | 0 | 2 | 2 | 4 | 4 | 2 | 3 | 6 | 3 | 6 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1 | 2 | 0 | 0 | 2 | 2 | 2 | 1 | 1 | 1 | 1 | 2 | 4 | 2 | 5 | 6 | 9 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 2 | 3 | 5 | 1 | 3 | 5 | 4 | 4 | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 3 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 4 | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 3 | 0 | 2 | 0 | 3 | 1 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 2 | 2 | 1 | 5 | 1 | 2 | 2 | 0 | 8 | 6
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 2 | 1 | 1 | 3 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 2 | 1 | 3 | 2 | 2
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 4 | 0 | 4 | 2 | 4 | 1 | 3 | 6 | 4
Immune effector cell-associated neurotoxicity syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 1 | 0 | 0 | 1 | 0 | 4 | 3
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 2 | 0 | 1 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 0 | 2 | 3 | 3 | 3
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 1 | 4 | 2 | 4 | 2 | 3 | 5 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 6 | 0 | 1 | 2 | 1 | 4 | 7
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 1 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 0 | 2 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 2 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 1 | 2 | 0 | 3 | 3 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 2 | 3 | 4 | 4 | 3 | 6 | 0 | 7 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 1 | 2 | 2 | 0 | 2 | 1 | 5 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 1 | 1 | 2 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 1 | 0 | 2 | 0 | 4 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 2 | 0 | 2 | 1 | 0 | 5 | 2
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 2 | 2 | 3 | 2
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 2 | 2 | 1 | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-03-29): https://cdn.clinicaltrials.gov/large-docs/36/NCT03269136/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-14): https://cdn.clinicaltrials.gov/large-docs/36/NCT03269136/SAP_001.pdf